# An Open-Label, Parallel Study to Assess Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Nicotine Uptake During a 56-Day Switch to myblu<sup>TM</sup> e-Cigarettes in Adult Smokers

NCT# 04019626

Study SAP - 05 March 2020

#### Statistical Analysis Plan

An Open-Label, Parallel Study to Assess Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Nicotine Uptake During a 56-Day Switch to *my*blu<sup>TM</sup> e-Cigarettes in Adult Smokers

Protocol No: CA22747
Final Protocol Date: 28 January 2019

Amendment 1 Date: 23 April 2019 Protocol Amendment 2: 17 May 2019

Product Names: *my*blu<sup>™</sup> system with Tobacco Chill flavor Intense Liquidpod, 2.5% nicotine, *my*blu<sup>™</sup> system with Tobacco Chill flavor Intense Liquidpod, 4.0% nicotine, *my*blu<sup>™</sup> system with Honeymoon flavor Intense Liquidpod, 2.5% nicotine, *my*blu<sup>™</sup> system with Honeymoon flavor Intense Liquidpod, 4.0% nicotine

Project CA22747 Final Version 1.0 Date: 05 March 2020

Nerudia Ltd

# Statistical Analysis Plan Signature Page

Product Names: myblu<sup>TM</sup> system with Tobacco Chill flavor Intense Liquidpod, 2.5% nicotine, myblu<sup>TM</sup> system with Tobacco Chill flavor Intense Liquidpod, 4.0% nicotine, myblu<sup>TM</sup> system with Honeymoon flavor Intense Liquidpod, 2.5% nicotine, myblu<sup>TM</sup> system with Honeymoon flavor Intense Liquidpod, 4.0% nicotine

Protocol: CA22747

Study Title: An Open-Label, Parallel Study to Assess Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Nicotine Uptake During a 56-Day Switch to myblu<sup>TM</sup> c-Cigarettes in Adult Smokers

Issue Date: 05 March 2020



# **Table of Contents**

| 1. | INT | NTRODUCTION5 | | |
|---|---|---|---|---|
| 2. | | | ES AND ENDPOINTS | |
| | 2.1 | | | |
| | 2.2 | 3 | pints | |
| 3. | STU | DY DE | SIGN | 8 |
| 4. | | | | |
| т. | | | | |
| | | • | • | |
| | | | • • | |
| | 4.2 | | | |
| 5. | | | | |
| 6. | ANALYSIS OF STUDY ENDPOINTS | | | |
| | 0.1 | | | |
| | | | • | |
| | <del>_</del> | | | |
| | 0.2 | | | |
| | | | • | |
| | 6.1.2 Product Use and Compliance Data Summarization 6.2 Biomarkers of Exposure and Potential Harm 6.2.1 Biomarker Sample Collection 6.2.2 Biomarker Calculations Calculation of Urine Nicotine Equivalents Calculation of Total Mass Excreted | | | |
| | 2.1 Objectives 2.2 Endpoints STUDY DESIGN ANALYSIS POPULATIONS 4.1 Analysis Populations 4.1.1 Safety Population 4.1.2 Intent-to-Treat (ITT) Population 4.1.3 Per-Protocol Population (for the PK Sub-Study Evaluation) 4.1.4 Pharmacokinetic Population (for the PK Sub-Study Evaluation) 4.2 Preliminary Data and Interim Analysis PRODUCT DESCRIPTIONS ANALYSIS OF STUDY ENDPOINTS 6.1 Product Use and Compliance 6.1.1 Product Use and Compliance Assessments 6.1.2 Product Use and Compliance Data Summarization 6.2 Biomarkers of Exposure and Potential Harm 6.2.1 Biomarker Sample Collection 6.2.2 Biomarker Calculations Calculation of Urine Nicotine Equivalents Calculation of Total Mass Excreted Creatinine Adjustments 6.2.3 Biomarker Data Summarization 6.3 Physiologic Assessments 6.3.1 Physiologic Assessments 6.3.2 Data Summarization for Physiologic Assessments 6.4 Subjective Measures 6.4.1 Subjective Effects Questionnaire 6.4.2 Subjective Effects Data Summarization 6.5 Plasma Nicotine Pharmacokinetics 6.5.1 Measurements and Collection Schedule 6.5.2 Pharmacokinetic Concentrations 6.5.3 Plasma Nicotine Pharmacokinetic Parameters | | | |
| | 63 | | | |
| | 0.5 | | | |
| | 6.4 | | | |
| | | 3 | | |
| | | 6.4.2 | | |
| | 6.5 | Plasma Nicotine Pharmacokinetics | | |
| | | 6.5.1 | Measurements and Collection Schedule | 19 |
| | | 6.5.2 | Pharmacokinetic Concentrations | 19 |
| | | 6.5.3 | Plasma Nicotine Pharmacokinetic Parameters | |
| | | 6.5.4 | PK Data Summarization and Presentation | 21 |
| | 6.6 | Urge | to Smoke | 22 |

# Nerudia Ltd. *my*blu E-cigarettes

| | _ | 6.6.1 Urge to Smoke Parameters | 22 |
|---|---|---|---|
| | | 6.6.2 Urge to Smoke Data Summarization | |
| | 6.7 | Statistical Analyses | |
| | | 6.7.1 Statistical Analyses of Primary Endpoints | 23 |
| | | 6.7.2 Statistical Analyses of Secondary Endpoints | |
| 7. | SAFI | ETY | 24 |
| | 7.1 | Subject Discontinuation | |
| | 7.2 | Demographics | |
| | 7.3 | Smoking History | |
| | 7.4 | Adverse Events. | |
| | 7.5 | Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis) | 26 |
| | 7.6 | Vital Signs | 26 |
| | 7.7 | Electrocardiogram | 27 |
| | 7.8 | Concomitant Medications | 27 |
| | 7.9 | Physical Examination | 27 |
| | 7.10 | Exhaled CO | 27 |
| | 7.11 | Lung Function (Spirometry) | 28 |
| 8. | SUM | MARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 28 |
| 9. | SUMMARY TABLES AND FIGURES | | |
| | Section 14 Summary Tables and Figures | | |
| | | Section 16 Data Listings | |
| 10. | TAB | LE AND FIGURE SHELLS | 53 |
| | 10.1 | Figures Shells | 55 |
| | 10.2 | Post-Text Summary Tables Shells | 60 |
| 11 | LIST | TING SHELLS | 01 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from this study. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within protocol, after the locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by the Nerudia Ltd., will be considered out of scope and must be described in the CSR.

#### 2. OBJECTIVES AND ENDPOINTS

# 2.1 Objectives

#### Primary:

1. To assess the change-from-baseline differences in the primary tobacco-related biomarkers of exposure (BoE) following a 28-day use period of *my*blu<sup>TM</sup> electronic cigarettes (e-cigarettes) relative to smoking usual brand combustible cigarettes (UBCC).

### Secondary:

- 1. To assess the change-from-baseline differences in the primary tobacco-related BoE following a 56-day use period of *my*blu<sup>TM</sup> e-cigarettes relative to smoking usual brand combustible cigarettes.
- 2. To assess the change-from-baseline differences in the secondary tobacco-related BoE following 28-day and 56-day use periods of *my*blu<sup>TM</sup> e-cigarettes relative to smoking usual brand combustible cigarettes.
- 3. To characterize the change in the primary and secondary BoE and biomarkers of potential harm (BoPH) during a 56-day period of use of *my*blu<sup>TM</sup> e-cigarettes.
- 4. To assess the change-from-baseline differences in the primary and secondary tobaccorelated BoE between Day 28 and Day 56 in subjects using *my*blu<sup>TM</sup> e-cigarettes.
- 5. To assess change-from-baseline differences in the (BoPH following 28-day and 56-day use periods of *my*blu<sup>TM</sup> e-cigarettes relative to smoking usual brand combustible cigarettes.
- 6. To assess change-from-baseline differences in physiologic endpoints following 28-day and 56-day use periods of *my*blu<sup>TM</sup> e-cigarettes relative to smoking usual brand combustible cigarettes.
- 7. To assess elements of abuse liability, subjective effects, and perceptions associated with use of myblu<sup>TM</sup> e-cigarettes.
- 8. To characterize use of four *my*blu<sup>™</sup> e-liquids (Tobacco Chill and Honeymoon flavor Intense e-liquids, 2.5% and 4.0% nicotine) during a 56-day use period.

- 9. To characterize nicotine uptake from the *my*blu<sup>™</sup> e-cigarettes relative to an e-cigarette comparator (JUUL<sup>®</sup> Virginia Tobacco 5% nicotine) and usual brand combustible cigarettes.
- 10. To confirm the safety of myblu<sup>TM</sup> e-cigarettes during a 56-day use period.

# 2.2 Endpoints

# **Hypothesis:**

Switching from usual brand combustible cigarettes to a *my*blu<sup>TM</sup> e-cigarette will result in a significant decrease from baseline in the primary tobacco-related BoE following 28 days of use relative to the change associated with continuing to smoke combustible cigarettes. The hypothesis will be tested independently for each *my*blu<sup>TM</sup> e-liquid Product.

# **Primary Study Endpoints:**

# 1. Biomarkers of Exposure

| Biomarker | Matrix | <b>Chemical Constituent</b> |
|-----------------------------|--------|-----------------------------|
| Carboxyhemoglobin | Blood | Carbon monoxide (CO) |
| (COHb) | | |
| 4-(methylnitrosamino)-1-(3- | Urine | 4-(methylnitrosamino)-1-(3- |
| pyridyl)-1-butanol (NNAL) | | pyridyl)-1-butanone (NNK) |
| 3-hydroxypropylmercapturic | Urine | Acrolein |
| acid (3-HPMA) | | |
| S-phenyl mercapturic acid | Urine | Benzene |
| (S-PMA) | | |

# **Secondary Study Endpoints:**

#### 1. Biomarkers of Exposure

| Biomarker | Matrix | <b>Chemical Constituent</b> |
|-------------------------------|--------|-----------------------------|
| N-nitrosonornicotine (NNN) | Urine | NNN |
| 2-cyanoethyl-mercapturic acid | Urine | Acrylonitrile |
| (CEMA) | | |
| Hydroxyethyl mercapturic acid | Urine | Ethylene oxide |
| (HEMA) | | |
| 3-hydroxy-1- | Urine | Crotonaldehyde |
| methylpropylmercapturic acid | | |
| (HMPMA) | | |
| Monohydroxybutenylmercapturic | Urine | 1,3-butadiene |
| acid (MHBMA) | | |
| Hydroxypyrene (1-OHP) | Urine | Pyrene |
| o-toluidine (o-tol) | Urine | Toluidine |

| 3-hydroxybenzo[a]pyrene (3-OH | Urine | B[a]P |
|-------------------------------|-------|-------------|
| B[a]P) | | |
| 1-aminonaphthalene (1-AN) | Urine | Naphthalene |
| 2-aminonaphthalene (2-AN) | Urine | Naphthalene |
| Nicotine equivalents | Urine | Nicotine |

#### 2. Biomarkers of Potential Harm

| Biomarker | Matrix | Biological Effect |
|--------------------------------------|--------|---------------------|
| Soluble intracellular adhesion | Blood | Inflammation |
| molecule (sICAM) | | |
| White blood cells (WBCs) | Blood | Inflammation |
| High density lipoprotein cholesterol | Blood | Inflammation |
| (HDL-C) | | |
| Monocyte chemoattractant protein 1 | Blood | Inflammation |
| (MCP-1) | | |
| Type III isoprostane (8-epi- | Urine | Oxidative stress |
| prostaglandin $F_{2\alpha}$ ) | | |
| 11-dehydrothromboxane B <sub>2</sub> | Urine | Platelet activation |

#### 3. Physiological assessments

- Fractional concentration of exhaled nitric oxide (FeNO)
- Blood pressure
- Heart rate

#### 4. Subjective measures

- Penn State [Electronic] Cigarette Dependence Index (PSCDI, PSECDI)
- Cough Questionnaire
- Questionnaire of Smoking Urges-Brief (QSU-Brief)
- Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R)
- Product Evaluation Scale (PES)
- Product Liking Questionnaire
- Future Intent to Use Questionnaire
- Product and Health Effect Perceptions Questionnaire

#### 5. Product Use

Daily in-clinic product use documented by the clinic staff:

- Number of cigarettes smoked
- Number of *my*blu<sup>TM</sup> and JUUL® pods started
- myblu<sup>TM</sup> pod weight change (for pods used during the 24 hour urine collections)
- Day 3 and Day 29 product preference selection

Daily product use endpoints documented by subjects (Day 3 through study discharge on Day 57):

• Number of cigarettes smoked

- Number of *my*blu<sup>TM</sup> pods started
- Number of puffs from the *my*blu<sup>TM</sup> product daily (< or  $\ge$  50 puffs)

#### 6. Nicotine Pharmacokinetics Assessment

Product use during each product use session:

- Number of puffs taken
- myblu<sup>TM</sup> and JUUL<sup>®</sup> pod weight change

Pharmacokinetic (PK) parameters during each product use session:

- C<sub>max</sub>
- AUC<sub>0-t</sub>
- T<sub>max</sub>

#### 7. Urge to Smoke Parameters (during the *ad libitum* product use session)

- Maximum reduction from baseline score  $(E_{max R})$
- Time of the  $E_{max}$  R ( $TE_{max}$ )
- Area under the change from baseline "Urge to Smoke" visual analog scale (VAS) score versus time curve (AUEC <sub>BL</sub>)

# 8. Other Compliance Assessments

Exhaled CO and urine cotinine measurements will be used to confirm smoking/nicotine use status prior to Day 1 and to assess subject compliance with product assignment requirements thereafter.

#### 9. Safety Assessments

Safety endpoints will include physical examinations, vital signs, electrocardiograms (ECGs), clinical laboratory tests, lung function, pregnancy tests, AEs, and use of concomitant medications.

#### 3. STUDY DESIGN

This will be an open-label, partially-randomized, parallel-arm, multi-site study in healthy adult smokers, consisting of two parts – the main study and a PK sub-study.

<u>The main study</u> will assess BoE, BoPH, physiologic effects, and subjective effects with use of *my*blu<sup>TM</sup> e-cigarettes relative to continuing to smoke combustible cigarettes. To account for potential attrition, up to 160 subjects are planned to be randomized into the *my*blu<sup>TM</sup> arm (with up to 40 subjects intended to be assigned to each *my*blu<sup>TM</sup> e-liquid) and up to 40 subjects will be randomized into the continuesmoking arm.

Baseline study assessments will be made during use of subjects' usual brand combustible cigarettes during the initial test visit through the morning of Day 1. All subjects in the *my*blu<sup>TM</sup> and continue-smoking arms will return to the clinic site for test visits scheduled to occur on Days 14, 28, 42, and 56 for post-baseline study assessments, compliance checks, and product dispensing and return. The subset of

subjects participating in the PK sub-study (described below) will also complete selected biomarker assessments (NNAL, NNN, 3-HPMA, CEMA, HMPMA, S-PMA, nicotine equivalents) on Days 3 and 4.

Subjects randomized to the *my*blu<sup>TM</sup> arm will participate in an in-clinic product acclimation period from Days 1 to 3. The acclimation period will afford the subjects the opportunity to try each of the four *my*blu<sup>TM</sup> e-liquids in order to become accustomed to their use and to determine those that they would be willing to use during the study. Initial product assignment for each subject will be based on preference as a method to enhance compliance. To further improve compliance through Day 56, at the end of Test Visit 3, subjects using a *my*blu<sup>TM</sup> product may be allowed to choose to switch to the alternate nicotine strength of their current flavor, to switch to the alternate flavor with the same nicotine strength as their initial choice, or to continue using the same e-liquid selected initially. This method for initial flavor assignment and the opportunity to re-select after 28 days of use is based on natural experimentation that consumers experience when choosing an e-cigarette flavor.

The PK sub-study will assess nicotine uptake and urge to smoke from the myblu<sup>TM</sup> products relative to combustible cigarettes and an e-cigarette comparator (JUUL®). A subset of up to 20 subjects assigned to each of the myblu<sup>TM</sup> e-liquids, 20 subjects from the continue-smoking arm, and all 20 subjects in the JUUL® arm will participate. Subjects in the JUUL® arm will begin using the product after check-in (Day -2) for Test Visit 1 and will continue to use the product through discharge on Day 1 from the study following the PK assessment (subjects in the JUUL® arm will only participate in the PK sub-study). PK assessments will be preceded by a minimum 10-hour abstention from product use and will take place on Day 1 for the JUUL<sup>®</sup> and continue-smoking arms, and on Day 5 for the *my*blu<sup>TM</sup> arm. Product use for the PK assessments will consist of two sessions: 1) a fixed/controlled puffing session in the morning consisting of 10 puffs taken at 30 second intervals, with puffs 3 seconds in duration, and 2) an *ad libitum* use session beginning 6 hours after the start of the morning session and consisting of unlimited use of the e-cigarette product for 5 minutes or one cigarette, with no limits on puff duration or inter-puff interval. No product use of any kind will be allowed between the sessions. E-cigarette pods used for each session will be weighed before and after use to measure the amount of e-liquid used.

All product use during confinement will be documented by the clinic staff. Subjects in the *my*blu<sup>TM</sup> and continue-smoking arms will be required to self-report product use from Day 3 through discharge from the study.

Exhaled CO and urine cotinine measurements will be used to confirm smoking/nicotine use status prior to Day 1 and to assess subject compliance with product assignment requirements thereafter.

The clinic staff will contact all subjects via a telephone call approximately 14 days after discharge from the study (either as scheduled or after early termination) for reporting of AEs and use of concomitant medications.

Screening of subjects will occur within 28 days prior to prior to check-in (Day -2) for Test Visit 1. Screening safety evaluations will include a physical examination, vital signs, ECG, clinical laboratory tests (clinical chemistry, hematology, urinalysis, and serology), lung function, urine drug tests, urine cotinine tests, and alcohol breath tests, FSH tests (post-menopausal females) and serum and urine pregnancy tests (females only).

On-study safety evaluations will include a symptom-driven physical examinations, vital signs, ECG, clinical laboratory tests (clinical chemistry, hematology, and urinalysis), lung function, and urine pregnancy tests (females only).

AEs spontaneously reported by the subjects or observed by the Investigator or other study personnel will be documented and monitored from the time of first product use after successful completion of the check-in (Day -2) events for Test Visit 1 through the end of the Follow-up Period. Any prior and concomitant medications taken from 30 days prior to Screening through the Follow-up Period will also be recorded.

# **Product Use**

#### Baseline and Product Use Period 1 (Days -2 to 29, Test Visits 1-3):

Subjects who meet study requirements following screening will be scheduled to check in to the clinic for Test Visit 1 on Day -2 (check-in for JUUL® arm will be as early in the day as possible to maximize the time to use the product) and will remain in the clinic until completion of all study events. Subjects who fail the check-in requirements will be considered a "screen failure" and will be excluded from participation. For the *my*blu<sup>TM</sup> and continue-smoking arms, the Baseline Period will consist of the time between check-in and first product use on Day 1.

Following discharge from Test Visit 1 (Day 5), subjects in the *my*blu<sup>TM</sup> and continue-smoking arms will follow the product use requirements of their randomization arm and will report product use daily. All subjects in the *my*blu<sup>TM</sup> and continue-smoking arms will be required to present to the clinic site on Day 14 and Day 28 (each ± 2 days) for Test Visits 2 and 3, respectively. Test Visit 2 will be ambulatory and primarily for the return and dispensing of test products for the *my*blu<sup>TM</sup> arm and for compliance and safety checks for both study arms. Test Visit 3 (Days 28 and 29) will be for these purposes in addition to completion of the endpoint assessments during confinement.

#### Product Use Period 2 (Days 30 to 57, Test Visits 4 and 5):

Following discharge from Test Visit 3, subjects in the *my*blu<sup>™</sup> and continue-smoking arms will follow the product use requirements of their randomization arm and will report product use daily. All subjects in both arms will be required to present to the

clinic site on Day 42 and Day 56 (each  $\pm$  2 days) for Test Visits 4 and 5, respectively. Test Visit 4 will be ambulatory and primarily for the return and dispensing of test products for the myblu<sup>TM</sup> arm and for compliance and safety checks for both study arms. Test Visit 5 will be for these purposes in addition to completion of the endpoint assessments during confinement. Subjects will be discharged from the clinical portion of the study at the end of Test Visit 5.

#### 4. ANALYSIS POPULATIONS

#### 4.1 Analysis Populations

#### 4.1.1 Safety Population

The safety population will include all subjects with at least one reported product use from Day -1.

# 4.1.2 Intent-to-Treat (ITT) Population

The ITT population will consist of randomized subjects in the main study with at least one documented product-use experience from Day 1, irrespective of their compliance of the product-use to which they were randomized.

### 4.1.3 Per-Protocol Population

The PP population (main study) is a subset of the ITT population who meet the requirements below. Separate populations for Product Use Period 1 (PP28/29) and Product Use Period 2 (PP56/57) will be established based on data collected during each of those periods.

The PP population will be used (in addition to the ITT population) only in the analysis of primary biomarkers of exposure (COHb in plasma and NNAL, 3-HPMA, and S-PMA in urine) and in the product use analysis.

#### myblu<sup>TM</sup> and continue-smoking arms

- Have no protocol deviations significantly impacting the integrity of the analysis or interpretation of the individual endpoint under consideration (e.g., compromised urine samples, use of prohibited medications impacting the endpoint)
- Have a daily product use response rate of at least 70% during the product use period
- Have a positive urine cotinine test at each scheduled assessment.

#### myblu<sup>TM</sup> arm

• Self-report reducing cigarette consumption by at least 90% of that reported at baseline

- Have exhaled CO values  $\leq 8$  ppm at each scheduled post-baseline assessment
- Have post-baseline urine NNAL values reduced by  $\geq 75\%$  from baseline.

# 4.1.4 Pharmacokinetic Population (for the PK Sub-Study Evaluations)

The PK population for each product use session will include subjects who used a product and have evaluable PK profiles. This population will include approximately half (up to 20 out of 40) of the subjects from each of the four *my*blu<sup>TM</sup> arms and from the Cigarette arm, plus all subjects (20) from the JUUL® arm. The sub-study will therefore include approximately 120 subjects, of which 100 subjects would also participate in the main study and 20 subjects (the JUUL® arm) exclusively in the substudy.

#### 4.2 Preliminary Data and Interim Analysis

Preliminary analyses may be performed, as judged applicable.

#### 5. PRODUCT DESCRIPTIONS

All subjects will be required to provide a sufficient supply of their usual brand combustible cigarettes to the study site for use on Day 1.

Each subject's usual brand information, including Universal Product Code (UPC) number, will be documented.

The following investigational products will be used during the study:

- myblu<sup>TM</sup> system with Tobacco Chill flavor Intense Liquidpod, 2.5% nicotine
- myblu<sup>TM</sup> system with Tobacco Chill flavor Intense Liquidpod, 4.0% nicotine
- myblu<sup>TM</sup> system with Honeymoon flavor Intense Liquidpod, 2.5% nicotine
- myblu<sup>TM</sup> system with Honeymoon flavor Intense Liquidpod, 4.0% nicotine

Each blu e-liquid contains a mixture of glycerin, propylene glycol, nicotine, and a proprietary blend of flavors.

The following comparator products will be used during the study:

- Subject's usual brand combustible cigarette
- JUUL® system with Virginia Tobacco Flavor JUULpod, 5.0% nicotine

In the CSR text and table headings, product use will be referred to by the short descriptions; the 6 products referred to as Products A-F and table footers by the long description in the following table:

**Table 5.1. Product Description** 

| Arm | Products | oducts Short Description | | Long Description |
|---|---|---|---|---|
| | A | myblu™ Tobacco<br>Chill 2.5% | e-cigarette | <i>my</i> blu <sup>™</sup> closed system with CF<br>Cosmic Fog Tobacco Chill flavor,<br>nicotine salt liquid 2.5 % |
| A | В | myblu™ Tobacco<br>Chill 4.0% | e-cigarette | myblu™ closed system with CF<br>Cosmic Fog Tobacco Chill flavor,<br>nicotine salt liquid 4.0% |
| | С | <i>my</i> blu™ Honeymoon 2.5% | e-cigarette | <i>my</i> blu <sup>™</sup> closed system with CF<br>Cosmic Fog Honeymoon flavor,<br>nicotine salt liquid 2.5 % |
| | D | <i>my</i> blu™ Honeymoon 4.0% | e-cigarette | <i>my</i> blu <sup>™</sup> closed system with CF<br>Cosmic Fog Honeymoon flavor,<br>nicotine salt liquid 4.0% |
| R F Cigarette | | combustibl<br>e cigarette | Subject's usual brand combustible cigarette | |
| С | C F JUUL® e-c | | e-cigarette | JUUL® system with Virginia<br>Tobacco Flavor JUULpod, 5.0%<br>nicotine |

#### 6. ANALYSIS OF STUDY ENDPOINTS

# 6.1 Product Use and Compliance

#### **6.1.1 Product Use and Compliance Assessments**

#### myblu<sup>TM</sup> Product Use

Following product training on Day 1, subjects will use each of the four test products individually for approximately 2 hours each, with the order of use selected by the subject. Following the last 2-hour period, subjects may choose any of the e-liquids freely through 23:00 on Day 2. At 20:00 on Day 2, subjects will complete the *my*blu<sup>TM</sup> Product Preference Questionnaire. Initial product assignment for each subject will be made by the study statistician or designee. Beginning on the morning of Day 3, subjects will use the assigned e-liquid through Day 28 and will be given the opportunity at Visit 3 to switch to the alternate nicotine strength of their current flavor, to switch to the alternate flavor with the same nicotine strength as their initial choice, or to continue using the same e-liquid selected initially through Day 57 (Visit 5, last study day). Each day from Day 3 through discharge from the study on Day 57, subjects randomized to the *my*blu<sup>TM</sup> arm will self report their product use via a text message system (Medquest).

Subjects participating in the PK sub-study will continue to use the assigned product through the evening of Day 4. All pods used during the 24-hour urine collections will be weighed within 24 hours before and after use, with the weights documented. On Test Visit 3 (Day 28) and Test Visit 5 (Day 56) as well, all pods used during the 24-hour urine collections will be weighed within 24 hours before and after use, with the weights documented.

#### **Usual Brand Cigarette Use**

Subjects randomized to the continue-smoking arm will smoke their usual brand cigarettes at home and throughout each confinement visit, and will self-report the number of cigarettes smoked each day from Day 3 through discharge from the study via a text message system.

# JUUL® Product Use

Subjects in the JUUL® arm will begin using the product following the demonstration and training on Day -2 and will continue to use the product through 23:00 on Day -1.

#### **Product Use Compliance**

Subject self-reported product use will be used as a measure of compliance. The clinic staff will monitor the frequency with which subjects complete the daily product use entries leading up to each Test Visits 2 through 5.

Biochemical verification of compliance will also be performed. Exhaled CO and urine cotinine will be used as methods of verifying compliance in real-time.

NNAL is a tobacco-specific nitrosamine with a longer half-life than CO, thus may provide an estimate of compliance over a long period of time by comparison of the post-baseline values to the baseline values. As this will be measured in a bioanalytical assay, real-time monitoring will not be possible and the verification will be completed at the end of the study.

NNAL will be considered as an additional exploratory variable for compliance.

#### 6.1.2 Product Use and Compliance Data Summarization

The following product use variables will be determined:

#### PK Sub-Study

- Number of puffs taken during each controlled and ad libitum product use session
- myblu<sup>TM</sup> and JUUL<sup>®</sup> pod weight change (only on Day 5 or Day 1, respectively)

#### In-clinic

- Number of cigarettes smoked
- Number of *my*blu<sup>TM</sup> pods started

- myblu<sup>TM</sup> pod weight change (for pods used during the 24 hour urine collections)
- Day 3 and Day 29 product preference selection (a listing)

# Self report

- Number of cigarettes smoked (*my*blu<sup>TM</sup> and cigarette arms)
- Number of *my*blu<sup>TM</sup> pods started (*my*blu arm)
- > 50 puffs taken from of myblu<sup>TM</sup> product (Y/N) (myblu<sup>TM</sup> arm)

#### Compliance

- $\geq$  90% reduction of cigarette use from baseline (*my*blu<sup>TM</sup> arm)
- $\geq 70\%$  daily product use reporting (yes/no) all cohorts
- Measured eCO (≤8 ppm) all cohorts
- $\geq 75\%$  reduction in post-baseline urine NNAL from baseline (*my*blu<sup>TM</sup> arm)
- Urine cotinine (yes/no) all cohorts

All product use data (including the number of puffs and including the PK product use sessions) and compliance variables will be summarized by study product using descriptive statistics (by time point, day, and product use session as appropriate) but no statistical comparisons will be made. The difference in weight before and after use of each e-cigarette (Products A to D and Product F) will be summarized.

<u>For the PK sub-study</u>, the number of puffs and the difference in weight before and after use of each e-cigarette will also be summarized.

The level of precision for each statistic will be presented as follows:

- minimum/maximum in same precision as the data,
- arithmetic mean/median in one more level of precision than minimum/maximum,
- SD in one more level of precision than mean/median,
- n will be presented as an integer,
- arithmetic CV% will be presented to 1 decimal point, and

# 6.2 Biomarkers of Exposure and Potential Harm

#### **6.2.1** Biomarker Sample Collection

#### **Blood Biomarker Sample Collection**

Blood samples for COHb in whole blood (2 x 4 mL), sICAM in plasma (1 x 4 mL), WBCs in whole blood (measured in hematology sample), HDL-C in serum (1 x 3.5 mL), MCP-1 in serum (1 x 3.5 mL), and serum for bio-banking (up to 17 mL) will be collected during Test Visit 1 (on Days -2, and -1), Test Visit 3 (Days 28 and 29), and Test Visit 5 (Days 56 and 57). Samples for COHb will be collected in the afternoon

and samples for the other biomarkers and bio-banking will be collected following an overnight ITTt of at least 8 hours.

### **Urine Biomarker Sample Collection**

24-hour urine collections for biomarker measurements (NNAL, 3-HPMA, S-PMA, NNN, CEMA, HEMA, HMPMA, MHBMA, 1-OHP, (-tol, 3-OH B[a]P, 1-AN, 2-AN, nicotine equivalents, 8-epi-prostaglandin  $F_{2\alpha}$ , and 11-dehydrothromboxane  $B_2$ ) will take place, as applicable, during Test Visit 1 (on Days -2, -1, 3, and 4), Test Visit 3 (Days 28 and 29), and Test Visit 5 (Days 56 and 57). Each 24-hour urine collection will begin at a time following check-in and will end at the same time  $\pm$  30 minutes the following day.

Subjects will be instructed to attempt to void prior to the beginning and at the end of each interval. All urine must be collected during the entire 24-hour interval. The start and stop time of each 24-hour interval and the total weight of the collection will be documented. The weight of the 24-hour urine collection containers will be documented prior to the collection (tare weight) and following completion of the collection.

Collections for each subject will be pooled into one labeled container throughout the interval and the total weight (g) will be recorded at the end of the 24-hour interval. Any missed voids will be documented, including the reason for missing.

#### 6.2.2 Biomarker Calculations

#### **Calculation of Urine Nicotine Equivalents**

Nicotine equivalents will be calculated as the molar sum of nicotine and 5 major nicotine metabolites. Values of individual components reported as below the limit of quantitation (BLQ) will be set to one-half of the limit of quantitation in the calculation below. Missing urine data will not be imputed.

Nicotine equivalents ( $\mu$ g/mL) = (nicotine [ng/mL]/162.23 [mg/mmol] + nicotine-gluc (ng/mL)/338.36 [mg/mmol] + cotinine [ng/mL]/176.22 [mg/mmol] + cotinine-gluc [ng/mL]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [ng/mL]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [ng/mL]/368.34 [mg/mmol]) x 162.23 (mg/mmol) x 1  $\mu$ g/1000 ng

#### **Calculation of Total Mass Excreted**

Urine biomarker concentrations will be converted into biomarker quantities excreted in 24 hours by multiplying the measured concentration by the total weight (i.e., 1 kilogram = 1 liter) of urine produced by the subject during the 24-hour period.

#### **Creatinine Adjustments**

Urine creatinine will be measured and used to adjust the values of the primary and secondary urine BoPH and BoE as follows.

Biomarker =  $\underline{\text{Biomarker (units) x } 100}$ (unit/g creatinine) =  $\underline{\text{creatinine (mg/dL)}}$ 

#### 6.2.3 Biomarker Data Summarization

Biomarker concentrations reported as below the limit of quantitation will be reported as "BLQ" in the listings and set to one-half of the limit of quantitation for summarization and statistical analysis.

The following variables will be determined and summarized for each urine biomarker.

- Measured concentration
- Total biomarker mass excreted per 24 hours
- Creatinine-adjusted excretion level

Absolute and percent change-from-baseline will be determined for the mass excreted and creatinine-adjusted values. The total urine biomarker mass excreted per 24 hours change-from-baseline value will be used in the statistical analysis.

Data will be listed by subject, product, and visit or day (and time point as applicable) and summarized by product and visit or day (and time point as necessary). Absolute and percent change-from-baseline values, and absolute and percent differences between Test Visits 3 and 5 (Days 28 and 56, respectively), will also be listed and summarized where indicated.

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be presented. Figures will be used to display the data graphically as applicable. All data summarizations and figures will be generated using the ITT population. In addition, PP population will also be used for the primary biomarkers only: COHb in plasma and NNAL, 3-HPMA, and S-PMA in urine. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in Section 6.7.

# 6.3 Physiologic Assessments

#### **6.3.1** Physiologic Assessments and Visits

Test Visit 1, 3, and 5 check-in blood pressure (systolic and diastolic) and heart rate measurements will be assessed for physiologic assessment purposes.

#### 6.3.2 Data Summarization for Physiologic Assessments

Data will be listed by subject, product, and visit or day (and time point as applicable) and summarized by product and visit or day (and time point as necessary). Absolute and percent change-from-baseline values, and absolute and percent differences between Test Visits 3 and 5, will also be listed and summarized, as applicable.

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be used for continuous data variables and frequency counts (number of observations and percentage) for categorical data variables.

Figures may be used to display the data graphically, as applicable. All data summarizations including figures will be generated using the ITT population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in Section 6.7.

# 6.4 Subjective Measures

#### **6.4.1** Subjective Effects Questionnaire

The PSCDI/PSECDI, Cough Questionnaire, QSU-Brief, MTWS-R, PES, Product Liking Questionnaire, Future Intent to Use Questionnaire, and Product and Health Effect Perceptions Questionnaire will be completed during Test Visit 1 (Day -2), Test Visit 3 (Day 28), and Test Visit 5 (Day 56), as applicable, using an electronic device. The QSU-Brief, MTWS-R, PES, and Product Liking Questionnaire will also be completed on Day 3 (Visit 1).

# 6.4.2 Subjective Effects Data Summarization

The following total scores, factor scores, and subscales will be calculated and summarized. For questionnaires without total scores, factor scores, or subscales (Cough Questionnaire, Product Liking Questionnaire, Future Intent to Use Questionnaire, and Product and Health Effect Perceptions Questionnaire), each item on the subjective measures questionnaires will be summarized.

- PSCDI/PSECDI total score
- MTWS-R total score
- QSU-brief factor scores:
  - Factor 1 (anticipation of pleasure from smoking) average of items 1, 3, 6, 7, and 10
  - o Factor 2 (relief of nicotine withdrawal) average of items 2, 4, 5, 8, and 9
- PES subscales:

- o Satisfaction average of items 1, 2, 3, and 12
- Psychological reward average of items 4 through 8
- o Aversion average of items 9, 10, 16, and 18
- o Relief average of items 11, 13, 14, 15, and reversed for item 20
- o Items 17, 19, 21 will be summarized as individual item scores.

Data will be listed by subject, product, and visit or day (and time point as applicable) and summarized by product and visit or day (and time point as necessary). Absolute and percent change-from-baseline values, and absolute and percent differences between Test Visits 3 and 5, will also be listed and summarized, as applicable. Baseline is the last no-missing observation collected prior to Day 1 product use.

Descriptive statistics (number of observations, mean, median, standard deviation, standard error of the mean, CV%, minimum, and maximum) will be used for continuous data variables and frequency counts (number of observations and percentage) for categorical data variables.

Figures may be used to display the data graphically, as applicable. All data summarizations including figures will be generated using the ITT population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in Section 6.7.

#### 6.5 Plasma Nicotine Pharmacokinetics

#### 6.5.1 Measurements and Collection Schedule

PK assessments will take place on Day 1 for the JUUL® and continue-smoking arms, and on Day 5 for the *my*blu<sup>TM</sup> arm. A 4 mL blood sample for plasma nicotine analysis will be drawn into a plastic K2-EDTA (lavender top) vacutainer tube approximately 5 minutes prior to and at 3, 5, 7, 10, 12, 15, 20, 30, 60, 120 and 180 minutes following the start of each product use episode (fixed/controlled and *ad libitum*).

#### 6.5.2 Pharmacokinetic Concentrations

Plasma concentrations of nicotine as determined at the collection times described in Section 6.2.1 will be used for the calculation of the plasma nicotine PK parameters.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there are any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. All deviations and excluded data will be provided and discussed in the CSR.

#### 6.5.3 Plasma Nicotine Pharmacokinetic Parameters

The appropriate noncompartmental PK parameters will be calculated for each product use episode (controlled and *ad libitum*) from the baseline adjusted plasma nicotine concentration-time data using Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. The calculation of the actual time for nicotine will be in respect to the start of product use episodes on Day 1 for the JUUL<sup>®</sup> and continue-smoking arms, and on Day 5 for the *my*blu<sup>TM</sup> arm. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated (Baseline Adjusted)

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t | Area under the nicotine concentration-time curve from time 0 (defined as the start of product use) to 180 minutes (or the last quantifiable concentration during the interval) | Calculated using the<br>Linear Trapezoidal with<br>Linear Interpolation<br>Method |
| Cmax | Maximum measured plasma concentration over the duration of the measurement interval | Taken directly from bioanalytical data |
| Tmax | Time to reach the maximum measured plasma concentration over the duration of the measurement interval. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value. | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |

Pharmacokinetic parameters will not be calculated for subjects with less than 3 consecutive post-product use time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the descriptive statistics.

For the calculation of the PK parameters, plasma concentrations that are BLQ will be set to one-half of the LLOQ for the calculation of descriptive statistics of unadjusted plasma nicotine concentrations. Baseline adjustments (pre-product use) will be performed for calculation of PK parameters. The values used for all pre-product use adjustments is the plasma nicotine concentration value obtained before the first product use on Day 1-6 and the adjustment will be subject-specific.

Baseline-adjustment method: For each PK profile, the pre-product administration nicotine concentration value for each subject will be subtracted from each nicotine concentration obtained after test product administration on that day/episode using the following equation:

$$C_t = C_{t \text{ uncorrected}} - [C_0 \cdot e^{-Kel \cdot t1}]$$

Where:

 $C_t$  = Corrected concentration.

 $C_{t \text{ uncorrected}}$  = the uncorrected concentration.

 $C_0$  = the pre-product administration concentration.

$$Kel = \frac{\ln(2)}{t_{1/2}}$$

Where t1/2 is 2.0 hours for all subjects (estimated nicotine half-life)

t = actual sampling time since product administration.

t1 = actual sampling time since pre-product administration sampling.

After correction for pre-product administration values, some concentrations may be below the lower limit of quantitation and some may be negative values. Negative values will be assigned a value of zero in the analyses and all other values obtained will be reported as is even if these values are BLQ.

#### 6.5.4 PK Data Summarization and Presentation

All nicotine PK concentrations and/or PK parameters descriptive statistics will be generated using SAS® version 9.4 or higher.

The plasma concentrations of nicotine will be listed and summarized by product, product use episode, and time point for all subjects in the PK Population. Unadjusted and baseline adjusted plasma concentrations of nicotine will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including number of observations (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), minimum, median, maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semilog scales. Linear mean plots will be presented with and without SD.

Plasma nicotine PK parameters will be listed and summarized by product, product use episode, and time point for all subjects in the PK Population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax, which will be presented with 2 decimal places. Summary statistics (n, arithmetic mean, geometric mean, SD, CV%, geometric CV% (Geom CV%), minimum, median, maximum), will be calculated for plasma nicotine PK parameters AUC0-t, Cmax, and Tmax. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and/or parameter output,
- mean/geometric mean/median in one more level of precision than minimum/maximum,
- SD in one more level of precision than mean/median,
- n will be presented as an integer, and
- CV% and Geom CV% will be presented to the nearest tenth.

Statistical analyses will be performed using SAS and are described in Section 6.7.

# 6.6 Urge to Smoke

#### **6.6.1** Urge to Smoke Parameters

Urge to smoke will be assessed using a 100 mm VAS approximately 10 minutes prior to and within approximately 30 seconds prior to the scheduled blood draws at 5, 10, 15, 30, 60, and 120 minutes following the start of the *ad libitum* product use session.

The following parameters will be calculated for the urge to smoke assessments performed during the PK assessments.

 $E_{max\_R}$  The maximum reduction from baseline VAS score (VASpre-use – VASpost-use).

TE<sub>max</sub> Time of the  $E_{max\_R}$ . If the maximum value occurred at more than one time point,  $TE_{max}$  will be defined as the first time point with this value.

AUEC\_0-120\_R The area under the reduction from baseline "Urge to Smoke" VAS score (VASpre-use – VASpost-use) versus time curve from 0 to 120 minutes, calculated using the linear trapezoidal method with linear interpolation using actual sample times

#### 6.6.2 Urge to Smoke Data Summarization

Data will be listed by subject, product, and day (and time point as applicable) and summarized by product and visit (and time point as applicable).

Descriptive statistics (number of observations, mean, median, standard deviation, minimum, and maximum) will be used for continuous data variables.

Figures may be used to display the data graphically, as applicable. All data summarizations and figures will be generated using the PK Population. Data summarizations and statistical analyses will be performed using SAS procedures. Statistical analyses are described in Section 6.7.

#### 6.7 Statistical Analyses

# 6.7.1 Statistical Analyses of Primary Endpoints

# Statistical Analyses of Primary BoE (Day 28 only) (*my*blu<sup>TM</sup> Products Versus the Continue-smoking Arm)

Comparisons of the Day 28 primary BoE (COHb, NNAL, 3-HPMA, and S-PMA) change-from-baseline values between the continue-smoking arm and each *my*blu<sup>TM</sup> e-liquid product selected at Day 2 will be made using a linear mixed model ANOVA.

The ITT population will be used as the primary analysis population and an analysis using the PP population will be used as a supportive analysis.

The ANOVA model will include product arm, study day, and product arm by study day interaction as fixed effect and subject as a random effect. Least square means (LSMs) will be provided for each product arm at each study day. LSM differences, 95% confidence intervals of LSM differences, and p-values will be provided for the product arm comparisons at each study day. The comparisons of interest will include each of the *my*blu<sup>TM</sup> product arms compared to continue-smoking arm. The above statistical analyses will be performed using the following SAS codes.

Proc MIXED data=<>; Class subject arm day; Model dependent variable = arm day arm\*day/DDFM=KR; Random Subject; LSMeans arm day arm\*day/pdiff CL alpha=0.05; Run;

### 6.7.2 Statistical Analyses of Secondary Endpoints

Statistical Analyses of Primary BoE (Day 56 only), Secondary BoE, BoPH, Physiologic Endpoints, and Subjective Measure Endpoints (*my*blu<sup>TM</sup> Products Versus the Continue-smoking Arm)

An approach similar to that used for the primary endpoints will be used to make Day 28 and Day 56, as applicable, change-from-baseline comparisons between the *my*blu<sup>TM</sup> products and the continue-smoking arm for the applicable primary and secondary BoE, BoPH, physiologic endpoints, and subjective measure endpoints as described in the SAP. For the Day 56 analysis, the initial *my*blu<sup>TM</sup> flavor Product assignments for each subject will be maintained within the statistical model and a separate sensitivity analysis will be performed for subjects that do not switch flavors at Day 29.

The ITT population will be used for these analyses.

# Statistical Analyses of Primary BoE (Day 56 only) and Secondary BoE (Within *my*blu<sup>TM</sup> Products)

Comparisons of the primary and secondary BoE change-from-baseline values at each time point within the myblu<sup>TM</sup> products will also be made using a linear mixed model ANOVA.

# Statistical Analyses of Pharmacokinetics (*my*blu<sup>TM</sup> Products Versus the Continuesmoking arm or JUUL arm)

A linear mixed model ANOVA will be performed on the log-transformed nicotine PK parameters AUC and C<sub>max</sub> from each product use session (PK population). The model will include product arm as a fixed effect. Geometric LSMs will be provided for the PK parameters of Cmax and AUC by product arm. Geometric LSM ratio, 95% confidence intervals of geometric LSM ratio, and p-values will be provided for the product arm comparisons for Cmax and AUC. The comparisons of interest will include each of the *my*blu<sup>TM</sup> product arms compared to continue-smoking arm or JUUL arm. The above statistical analyses will be performed using the following SAS codes.

```
Proc MIXED data=<>;
Class subject arm;
Model LN_dependent variable = arm/DDFM=KR;
LSMeans arm/pdiff CL alpha=0.05;
Run;
```

Non-parametric analysis (Wilcoxon Rank Sum test) will be performed for the comparisons of  $T_{max}$  between test and reference products.

Similar methods will be used to compare the urge to smoke parameters.

#### 7. SAFETY

All case report form (CRF) data will be listed by subject and chronologically by assessment time points. This will include rechecks, unscheduled assessments, and early termination.

Applicable continuous variables will be summarized using n, arithmetic mean, SD, minimum, median, and maximum.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

# 7.1 Subject Discontinuation

Subjects will be summarized by number of subjects enrolled, randomized, completed, and discontinued the study with discontinuation reasons by randomized product arm and overall.

# 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) by randomized product arm and overall.

Frequency counts will be provided for categorical variables (race, ethnicity, and sex, and other characteristics) for each randomized product arm and overall.

#### 7.3 Smoking History

Descriptive statistics will be calculated for continuous variables (cigarettes smoked per day [CPD] and number of years smoked) by randomized product arm and overall.

Frequency counts will be provided for subject's usual brand for each randomized product arm and overall.

#### 7.4 Adverse Events

All adverse events (AEs) occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 21.0.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, product, severity, relationship to study product, and action; however, only product use-emergent AEs (PUEAEs) will be summarized.

A PUEAE is defined as an AE that is starting or worsening at the time of or after the first randomized study product use. Each PUEAE will be attributed to a study product based on the onset date and time of the AE.

If the onset time of an AE is missing and the onset date is the same as the first study product use date, then the AE will be considered product use emergent in the study product. If onset time of an AE is missing and the onset date does not fall on a study product use date, then the AE will be considered product use emergent for the last study product administered. If the onset date of an AE is missing, then the AE will be considered product use emergent, unless the onset date is known to have occurred within or between specific product use days.

PUEAEs will be tabulated by System Organ Class (SOC) and Preferred Term. Summary tables will include number of subjects reporting the AE and as percent of number of subjects used study product by product. The number of AEs will be tabulated in a similar manner. Tables which tabulate the number of PUEAEs by severity and relationship to study product will also be included.

In addition, adverse events occurred during baseline period on Day -2 and day -1 will be summarized separately.

Serious adverse events (SAEs), if present, will also be listed. Applicable narratives will be included in the CSR.

#### 7.5 Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis)

Serum Chemistry, hematology, and urinalysis samples will be collected at screening and check-in (Day -2) for all product arms. For *my*blu<sup>TM</sup> and continue-smoking arms, the clinical laboratory tests will also be performed at the end of Period 1 (Day 29) and the discharge from the study (Day 57, Period 2) or upon early termination.

Descriptive statistics will be reported for numeric clinical data and change from baseline by product arm and time point. Rechecked values prior to randomization will be used in calculating summary statistics. Baseline is the last non-missing value including recheck and unscheduled event before randomization (usually on Day -2 Check-in). Normal ranges will be listed.

Out of normal range and clinically significant laboratory values will be listed by subject. Results that are indicated as CS by the PI will be listed in the table.

A urine cotinine test will be completed at Screening and Check-in (Day -2) for all product arms. For *my*blu<sup>TM</sup> and continue-smoking arms, the urine cotinine test will also be performed on the first day of each Test Visit.

Urine drug tests and alcohol breath tests will be completed at Screening and Check-in (Day -2) for all product arms.

For females, serum pregnancy tests will be completed at Screening and urine pregnancy tests will be completed at Check-in for all product arms. For *my*blu<sup>™</sup> and continue-smoking arms, the urine pregnancy tests will also be performed on the first day of each Test Visit. Results for these tests will be listed as "Negative" or "Positive."

#### 7.6 Vital Signs

Vital signs (pulse and blood pressure) will be measured at Screening and Check-in for all product arms. For *my*blu<sup>TM</sup> and continue-smoking arms, the vital signs will also be performed at Day 5 and at Day 28, 29 (Period 1), and in Period 2 on Day 56 and at

the discharge from the study (Day 57) or upon early termination. For JUUL arm, the vital sign will be performed at Day 1 or upon early termination.

Descriptive statistics will be reported for vital sign measurements by product arm and time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

# 7.7 Electrocardiogram

A single 12-lead electrocardiogram (ECG) will be recorded at Screening for all product arms. For *my*blu<sup>TM</sup> and continue-smoking arms, the ECG will also be performed at the discharge from the study (Day 57) or upon early termination. For JUUL arm, the ECG will be performed at Day 1 and upon early termination.

Descriptive statistics will be reported for ECG parameters by product arm and time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

ECG results will be listed by subject.

#### 7.8 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Drug Dictionary Version 01MAR2018 and listed by subject.

#### 7.9 Physical Examination

Full physical examinations will be performed at Screening. For *my*blu<sup>™</sup> and continue-smoking arms, symptom driven physical examination will also be performed at Check-in (Day -2), Test Visit 1 discharge (Day 5) and at Day 28, 29 of Period 1, Day 56 of Period 2 and the discharge from the study (Day 57) or upon early termination. For JUUL arm, the symptom driven physical examination will be performed at Check-in (Day -2) and Day 1 or upon early termination.

Physical examinations will be listed by subject. Changes in physical examinations (if any) will be described in the text of the final report.

#### 7.10 Exhaled CO

Exhaled CO will be collected at Screening and Check-in (Day -2) for all product arms. For *my*blu<sup>TM</sup> and continue-smoking arms, exhaled CO will also be performed at Test Visit 1 discharge (Day 5) and at Day 28, 29 of Period 1, Day 56 of Period 2.

Descriptive statistics will be reported for exhaled CO by product arm and time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

Exhaled CO will be listed by subject.

# 7.11 Lung Function (Spirometry)

Subjects will undergo lung function testing at Screening to affirm eligibility (FEV<sub>1</sub>, FEV<sub>1</sub>:FVC ratio) and as a safety endpoint (FEV<sub>1</sub>, FVC, FEV<sub>1</sub>:FVC ratio, and forced expiratory flow (FEF)<sub>25-75%</sub>). For *my*blu<sup>TM</sup> and continue-smoking arms, spirometry will also be performed at the discharge from the study (Day 57) or upon early termination.

Descriptive statistics will be reported for measured and percent of predicted spirometry parameters by product arm and time point. Unscheduled events or rechecks post randomization will not be included in summaries. Similarly early termination results will not be included in summaries.

Spirometry results will be listed by subject.

#### 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.4 or higher.

#### **Section 14 Summary Tables and Figures**

The following is a list of table and figure titles that will be included in Section 14 of the report. Tables and figures may be renumbered as appropriate during the compilation of the report.

# 14.1 Demographic Data Summary Tables

| Table 14.1.1 | Summary of Disposition (Safety, ITT, and PP Populations) |
|--------------|-----------------------------------------------------------|
| Table 14.1.2 | Demographic Summary (Safety, ITT, and PP Populations) |
| Table 14.1.3 | Smoking History Summary (Safety, ITT, and PP Populations) |
| Table 14.1.4 | Summary of Disposition (PK Population) |
| Table 14.1.5 | Demographic Summary (PK Population) |
| Table 14.1.6 | Smoking History Summary (PK Population) |

# 14.2 Study Product Use, Biomarkers, Physiologic Assessments, Pharmacokinetics and Questionnaires Data Summary Tables and Figures

#### **14.2.1 Product Use Tables**

| 111211 1104400 | |
|---|---|
| Table 14.2.1.1 | Summary of In-Clinic Number of <i>my</i> blu <sup>™</sup> Pods Started by Product and Day (ITT) |
| Table 14.2.1.2 | Summary of In-Clinic Number of <i>my</i> blu <sup>™</sup> Pods Started by Product and Day (PP 28/29) |
| Table 14.2.1.3 | Summary of In-Clinic Number of <i>my</i> blu <sup>™</sup> Pods Started by Product and Day (PP 56/57) |
| Table 14.2.1.4 | Summary of In-Clinic Product Weight Changes by Product and Day (ITT) |
| Table 14.2.1.5 | Summary of In-Clinic Product Weight Changes by Product and Day (PP 28/29) |
| Table 14.2.1.6 | Summary of In-Clinic Product Weights Changes by Product and Day (PP 56/57) |
| Table 14.2.1.7 | Summary of In-Clinic Number of Cigarettes Smoked by Product and Day (ITT) |
| Table 14.2.1.8 | Summary of In-Clinic Number of Cigarettes Smoked Started by Product and Day (PP 28/29) |
| Table 14.2.1.9 | Summary of In-Clinic Number of Cigarettes Smoked by Product and Day (PP 56/57) |
| Table 14.2.1.10 | Summary of Self-Reported Number of <i>my</i> blu <sup>TM</sup> Pods Started by Product and Day (ITT) |
| Table 14.2.1.11 | Summary of Self-Reported Number of <i>my</i> blu <sup>TM</sup> Pods Started by Product and Day (PP 28/29) |
| Table 14.2.1.12 | Summary of Self-Reported Number of <i>my</i> blu <sup>TM</sup> Pods Started by Product and Day (PP 56/57) |
| Table 14.2.1.13 | Frequency of Self-Reported Number of Puffs Taken From $my$ blu <sup>TM</sup> product (>= 50) by Product and Day (ITT) |
| Table 14.2.1.14 | Frequency of Self-Reported Number of Puffs Taken From <i>my</i> blu <sup>TM</sup> product (>= 50) by Product Day (PP 28/29) |
| Table 14.2.1.15 | Frequency of Self-Reported Number of Puffs Taken From <i>my</i> blu <sup>TM</sup> product (>= 50) by Product and Day (PP 56/57) |

| Nerudia Ltd. | | |
|---|---|---|
| myblu E-cigarettes Clinical Study Report No. CA22747 | | |
| | Table 14.2.1.16 | Summary of Self-Reported Number of Cigarettes Smoked by Product and Day (ITT) |
| | Table 14.2.1.17 | Summary of Self-Reported Number of Cigarettes Smoked by Product and Day (PP 28/29) |
| | Table 14.2.1.18 | Summary of Self-Reported Number of Cigarettes Smoked by Product and Day (PP 56/57) |
| | Table 14.2.1.19 | Summary of Self-Reported Product Use by Product and Product Use Period (ITT) |
| | Table 14.2.1.20 | Summary of Self-Reported Product Use by Product and Product Use Period (PP 28/29) |
| | Table 14.2.1.21 | Summary of Self-Reported Product Use by Product and Product Use Period (PP 56/57) |
| | 14.2.2 Biomark | er Tables |
| | 14.2.2.1 Blood C | COHb |
| | Table 14.2.2.1.1. | Summary of Whole Blood COHb by Study Product and Study Day (ITT Population) |
| | Table 14.2.2.1.1. | Summary of Whole Blood COHb Change From Baseline by Study Product and Study Day (ITT Population) |
| | Table 14.2.2.1.1. | Summary of Whole Blood COHb Percent Change From Baseline by Study Product and Study Day (ITT Population) |
| | Table 14.2.2.1.1. | Summary of Whole Blood COHb by Study Product and Study Day (PP Population) |
| | Table 14.2.2.1.1. | Summary of Whole Blood COHb Change From<br>Baseline by Study Product and Study Day (PP<br>Population) |
| | Table 14.2.2.1.1. | 6 Summary of Whole Blood COHb Percent Change From Baseline by Study Product and Study Day (PP Population) |
| | Table 14.2.2.1.2. | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between <i>my</i> blu <sup>TM</sup> and Continuous<br>Smoking by Study Day (ITT Population) |
| | Table 14.2.2.1.2. | 2 Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between <i>my</i> blu <sup>TM</sup> and Continuous<br>Smoking by Study Day (PP Population) |
| | Table 14.2.2.1.3. | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between Day 28 and Day 56 in the<br><i>my</i> blu <sup>TM</sup> Groups (ITT Population) |

| inical Study Report No. | CAZZITI |
|---|---|
| Table 14.2.2.1.3.2 | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between Day 28 and Day 56 in the<br><i>my</i> blu <sup>TM</sup> Groups (PP Day56/57 Population) |
| Table 14.2.2.1.3.3 | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between Day 28 and Day 56 in the<br><i>my</i> blu <sup>TM</sup> Groups (PP Day56/57 Population – Sensitivity<br>Analysis) |
| Table 14.2.2.1.4.1 | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between <i>my</i> blu <sup>TM</sup> Groups by Study Day<br>(ITT Population) |
| Table 14.2.2.1.4.2 | Statistical Comparison of Whole Blood COHb Change<br>From Baseline Between <i>my</i> blu <sup>TM</sup> Groups by Study Day<br>(PP Population) |
| 14.2.2.2 Urine NNAL | |
| Table 14.2.2.2.1.1 | Summary of Urine NNAL 24-hour Amount Excreted by Study Product and Study Day (ITT Population) |
| Table 14.2.2.2.1.2 | Summary of Urine NNAL Amount Excreted Change<br>From Baseline by Study Product and Study Day (ITT<br>Population) |
| Table 14.2.2.2.1.3 | Summary of Urine NNAL Amount Excreted Percent<br>Change From Baseline by Study Product and Study<br>Day (ITT Population) |
| Table 14.2.2.2.1.4 | Summary of Urine NNAL Adjusted for Urine Creatinine by Study Product and Study Day (ITT Population) |
| Table 14.2.2.2.1.5 | Summary of Urine NNAL Adjusted for Urine<br>Creatinine Change From Baseline by Study Product and<br>Study Day (ITT Population) |
| Table 14.2.2.2.1.6 | Summary of Urine NNAL Adjusted for Urine<br>Creatinine Percent Change From Baseline by Study<br>Product and Study Day (ITT Population) |
| Table 14.2.2.2.1.7 | Summary of Urine NNAL Amount Excreted by Study<br>Product and Study Day (PP Population) |
| Table 14.2.2.2.1.8 | Summary of Urine NNAL Amount Excreted Change<br>From Baseline by Study Product and Study Day (PP<br>Population) |
| Table 14.2.2.2.1.9 | Summary of Urine NNAL Amount Excreted Percent<br>Change From Baseline by Study Product and Study<br>Day (PP Population) |

| J -1 | |
|---|---|
| Table 14.2.2.2.1.10 | Summary of Urine NNAL Adjusted for Urine Creatinine by Study Product and Study Day (PP Population) |
| Table 14.2.2.2.1.11 | Summary of Urine NNAL Adjusted for Urine<br>Creatinine Change From Baseline by Study Product and<br>Study Day (PP Population) |
| Table 14.2.2.2.1.12 | Summary of Urine NNAL Adjusted for Urine<br>Creatinine Percent Change From Baseline by Study<br>Product and Study Day (PP Population) |
| Table 14.2.2.2.2.1 | Statistical Comparison of Urine NNAL 24-hour<br>Amount Excreted Change From Baseline Between<br><i>my</i> blu <sup>TM</sup> and Continuous Smoking by Study Day (ITT<br>Population) |
| Table 14.2.2.2.2.2.2 | Statistical Comparison of Urine NNAL 24-hour<br>Amount Excreted Change From Baseline Between<br><i>my</i> blu <sup>TM</sup> and Continuous Smoking by Study Day (PP<br>Day28/29 Population) |
| Table 14.2.2.2.2.3 | Statistical Comparison of Urine NNAL 24-hour<br>Amount Excreted Change From Baseline Between<br><i>my</i> blu <sup>TM</sup> and Continuous Smoking by Study Day (PP<br>Day56/57 Population) |
| Table 14.2.2.2.2.4 | Statistical Comparison of Urine NNAL 24-hour<br>Amount Excreted Change From Baseline Between<br><i>my</i> blu <sup>TM</sup> and Continuous Smoking by Study Day (PP<br>Day56/57 Population – Sensitivity Analysis) |

#### 14.2.2.3 Urine 3-HPMA

*Tables 14.2.2.3.1.1 through 14.2.2.3.2.2.4 will be generated for Urine 3-HPMA similar to Urine NNAL.* 

#### 14.2.2.4 Urine S-PMA

Tables 14.2.2.4.1.1 through 14.2.2.4.2.24 will be generated for Urine S-PMA similar to Urine NNAL.

#### 14.2.2.5 Urine NNN

Tables 14.2.2.5.1.1 through 14.2.2.5.2.2., as applicable (ITT population only), will be generated for Urine NNN similar to Urine NNAL.

#### **14.2.2.6 Urine CEMA**

Tables 14.2.2.6.1.1 through 14.2.2.6.2.2, as applicable (ITT population only), will be generated for Urine CEMA similar to Urine NNAL.

#### **14.2.2.7 Urine HEMA**

Tables 14.2.2.7.1.1 through 14.2.2.7.2.2.2, as applicable (ITT population only), will be generated for Urine HEMA similar to Urine NNAL.

#### **14.2.2.8 Urine HMPMA**

Tables 14.2.2.8.1.1 through 14.2.2.8.2.2., as applicable (ITT population only), will be generated for Urine HMPMA similar to Urine NNAL.

#### **14.2.2.9 Urine MHBMA**

Tables 14.2.2.9.1.1 through 14.2.2.9.2.2., as applicable (ITT population only), will be generated for Urine MHBMA similar to Urine NNAL.

#### 14.2.2.10 Urine 1-OHP

Tables 14.2.2.10.1.1 through 14.2.2.10.2.2.2, as applicable (ITT population only), will be generated for Urine 1-OHP similar to Urine NNAL.

#### 14.2.2.11 Urine o-tol

Tables 14.2.2.11.1.1 through 14.2.2.11.2.2.2, as applicable (ITT population only), will be generated for Urine o-tol similar to Urine NNAL.

# 14.2.2.12 Urine 3-OH B[a]P

Tables 14.2.2.12.1.1 through 14.2.2.12.2.2, as applicable (ITT population only), will be generated for Urine 3-OH B[a]P similar to Urine NNAL.

#### 14.2.2.13 Urine 1-AN

Tables 14.2.2.13.1.1 through 14.2.2.13.2.2.2, as applicable (ITT population only), will be generated for Urine 1-AN similar to Urine NNAL.

#### 14.2.2.14 Urine 2-AN

Tables 14.2.2.14.1.1 through 14.2.2.14.2.2.2, as applicable (ITT population only), will be generated for Urine 2-AN similar to Urine NNAL.

#### 14.2.2.15 Urine Nicotine Equivalents

Tables 14.2.2.15.1.1 through 14.2.2.15.2.2.2, as applicable (ITT population only), will be generated for Urine Nicotine Equivalents similar to Urine NNAL.

#### 14.2.2.16 Plasma sICAM

Tables 14.2.2.16.1.1 through 14.2.2.15.2.2.2, as applicable (ITT population only), will be generated for Plasma sICAM similar to Whole Blood COHb.

#### 14.2.2.17 WBCs

Tables 14.2.2.17.1.1 through 14.2.2.17.2.2.2, as applicable (ITT population only), will be generated for Whole Blood WBCs similar to Whole Blood COHb.

#### 14.2.2.18 Serum HDL-C

Tables 14.2.2.18.1.1 through 14.2.2.18.2.2.2, as applicable (ITT population only), will be generated for Serum HDL-C similar to Whole Blood COHb.

#### 14.2.2.19 Serum MCP-1

Tables 14.2.2.19.1.1 through 14.2.2.19.2.2.2, as applicable (ITT population only), will be generated for Serum MCP-1 similar to Whole Blood COHb.

# 14.2.2.20 Urine Type III isoprostane (8-epi-prostaglandin F2α)

Tables 14.2.2.20.1.1 through 14.2.2.20.2.2.2, as applicable (ITT population only), will be generated for Urine Type III isoprostane (8-epi-prostaglandin  $F2\alpha$ ) similar to Urine NNAL.

#### 14.2.2.21 Urine 11-dehydrothromboxane B2

Tables 14.2.2.21.1.1 through 14.2.2.21.2.2, as applicable (ITT population only), will be generated for Urine 11-dehydrothromboxane B2 similar to Urine NNAL.

#### 14.2.3 Physiologic Assessments Tables

#### 14.2.3.1 FeNO

Tables 14.2.3.1.1.1 through 14.2.3.1.2.2.2, as applicable (ITT population only), will be generated for FeNO similar to Whole Blood COHb.

#### 14.2.3.2 Systolic Blood Pressure

Tables 14.2.3.2.1.1 through 14.2.3.2.2.2, as applicable (ITT population only), will be generated for Systolic Blood Pressure similar to Whole Blood COHb.

#### 14.2.3.3 Diastolic Blood Pressure

Tables 14.2.3.3.1.1 through 14.2.3.3.2.2.2, as applicable (ITT population only), will be generated for Diastolic Blood Pressure similar to Whole Blood COHb.

# **14.2.3.4 Heart Rate**

Tables 14.2.3.4.1.1 through 14.2.3.4.2.2.2, as applicable (ITT population only), will be generated for Heart Rate similar to Whole Blood COHb.

| 14.2.4 | <b>Pharmacokinetics</b> | <b>Tables</b> |
|--------|-------------------------|---------------|

| 1 | Time of the contract of the co |
|---|---|
| Table 14.2.4.1.1.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following <i>myblu</i> <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product A) (PK Population) |
| Table 14.2.4.1.1.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product A) (PK Population) |
| Table 14.2.4.1.2.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Controlled Use (Product B) (PK Population) |
| Table 14.2.4.1.2.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product B) (PK Population) |
| Table 14.2.4.1.3.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product C) (PK Population) |
| Table 14.2.4.1.3.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product C) (PK Population) |
| Table 14.2.4.1.4.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Controlled Use (Product D) (PK Population) |
| Table 14.2.4.1.4.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product D) (PK Population) |
| inical Study Report 110. | C1122 ( ¬ ) |
|---|---|
| Table 14.2.4.1.5.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Subject's Usual Brand Combustible Cigarette Following Controlled Use (Product E) (PK Population) |
| Table 14.2.4.1.5.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Subject's Usual Brand Combustible Cigarette Following Ad Libitum Use (Product E) (PK Population) |
| Table 14.2.4.1.6.1 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Controlled Use (Product F) (PK Population) |
| Table 14.2.4.1.6.2 | Unadjusted Plasma Nicotine Concentrations (ng/mL) Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Ad Libitum Use (Product F) (PK Population) |
| Table 14.2.4.2.1.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product A) (PK Population) |
| Table 14.2.4.2.1.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product A) (PK Population) |
| Table 14.2.4.2.2.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Controlled Use (Product B) (PK Population) |
| Table 14.2.4.2.2.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product B) (PK Population) |
| Table 14.2.4.2.3.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product C) (PK Population) |
| Table 14.2.4.2.3.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid |

| | 2.5 % Following Ad Libitum Use (Product C) (PK Population) |
|---|---|
| Table 14.2.4.2.4.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Controlled Use (Product D) (PK Population) |
| Table 14.2.4.2.4.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product D) (PK Population) |
| Table 14.2.4.2.5.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Subject's Usual Brand Combustible Cigarette Following Controlled Use (Product E) (PK Population) |
| Table 14.2.4.2.5.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following Subject's Usual Brand Combustible Cigarette Following Ad Libitum Use (Product E) (PK Population) |
| Table 14.2.4.2.6.1 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Controlled Use (Product F) (PK Population) |
| Table 14.2.4.2.6.2 | Baseline-Adjusted Plasma Nicotine Concentrations (ng/mL) Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Ad Libitum Use (Product F) (PK Population) |
| Table 14.2.4.3.1.1 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product A) (PK Population) |
| Table 14.2.4.3.1.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu™ Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product A) (PK Population) |
| Table 14.2.4.3.2.1 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4 % Following Controlled Use (Product B) (PK Population) |
| Table 14.2.4.3.2.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic |

| | Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4 % Following Ad Libitum Use (Product B) (PK Population) |
|---|---|
| Table 14.2.4.3.3.1 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Controlled Use (Product C) (PK Population) |
| Table 14.2.4.3.3.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product C) (PK Population) |
| Table 14.2.4.3.4.1 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4 % Following Controlled Use (Product D) (PK Population) |
| Table 14.2.4.3.4.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4 % Following Ad Libitum Use (Product D) (PK Population) |
| Table 14.2.4.3.5.1 | Baseline-Adjusted Plasma Nicotine PK Parameters<br>Following Subject's Usual Brand Combustible<br>Cigarette Following Controlled Use (Product E) (PK<br>Population) |
| Table 14.2.4.3.5.2 | Baseline-Adjusted Plasma Nicotine PK Parameters<br>Following Subject's Usual Brand Combustible<br>Cigarette Following Ad Libitum Use (Product E) (PK<br>Population) |
| Table 14.2.4.3.6.1 | Baseline-Adjusted Plasma Nicotine PK Parameters<br>Following JUUL® System With Virginia Tobacco<br>Flavor JUUL Pod, 5.0% Nicotine Following Controlled<br>Use (Product F) (PK Population) |
| Table 14.2.4.3.6.2 | Baseline-Adjusted Plasma Nicotine PK Parameters Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Ad Libitum Use (Product F) (PK Population) |
| Table 14.2.4.4.1.1 | Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameters Between myblu <sup>TM</sup> and Continuous Smoking or JUUL Following Controlled Use (PK Population) |
| Table 14.2.4.4.1.2 | Statistical Comparisons of Baseline-Adjusted Plasma<br>Nicotine PK Parameters Between myblu <sup>TM</sup> and |

| J I | |
|---|---|
| | Continuous Smoking or JUUL Following Ad Libitum Use (PK Population) |
| Table 14.2.4.4.2.1 | Nonparametric Statistical Comparisons of Plasma<br>Nicotine PK Parameter Tmax Between myblu <sup>TM</sup> and<br>Continuous Smoking or JUUL Following Controlled<br>Use (PK Population) |
| Table 14.2.4.4.2.2 | Nonparametric Statistical Comparisons of Plasma<br>Nicotine PK Parameter Tmax Between myblu <sup>TM</sup> and<br>Continuous Smoking or JUUL 1 Following Ad Libitum<br>Use (PK Population) |
| 14.2.5 Urge to Smok | te Tables |
| Table 14.2.5.1 | Urge to Smoke VAS Score Following <i>my</i> blu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following <i>Ad Libitum</i> Use (Product A) (PK Population) |
| Table 14.2.5.2 | Urge to Smoke VAS Score Following myblu™ Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product B) (PK Population) |
| Table 14.2.5.3 | Urge to Smoke VAS Score Fol-lowing myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product C) (PK Population) |
| Table 14.2.5.4 | Urge to Smoke VAS Score Following myblu™ Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product D) (PK Population) |
| Table 14.2.5.5 | Urge to Smoke VAS Score Following Subject's Usual<br>Brand Combustible Cigarette Following Ad Libitum<br>Use (Product E) (PK Population) |
| Table 14.2.5.6 | Urge to Smoke VAS Score Following JUUL® System With Virginia Tobacco Flavor JUUL Pod, 5.0% Nicotine Following Ad Libitum Use (Product F) (PK Population) |
| Table 14.2.5.7 | Urge to Smoke VAS Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product A) (PK Population) |
| Table 14.2.5.8 | Urge to Smoke VAS Parameters Following myblu™ Closed System With CF Cosmic Fog Tobacco Chill Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product B) (PK Population) |

| Table 14.2.5.9 | Urge to Smoke VAS Parameters Following myblu <sup>TM</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 2.5 % Following Ad Libitum Use (Product C) (PK Population) |
|---|---|
| Table 14.2.5.10 | Urge to Smoke VAS Parameters Following myblu <sup>™</sup> Closed System With CF Cosmic Fog Honeymoon Flavor, Nicotine Salt Liquid 4.0% Following Ad Libitum Use (Product D) (PK Population) |
| Table 14.2.5.11 | Urge to Smoke VAS Parameters Following Subject's Usual Brand Combustible Cigarette Following Ad Libitum Use (Product E) (PK Population) |
| Table 14.2.5.12 | Urge to Smoke VAS Parameters Following JUUL®<br>System With Virginia Tobacco Flavor JUUL Pod, 5.0%<br>Nicotine Following Ad Libitum Use (Product F) (PK<br>Population) |
| Table 14.2.5.13 | Statistical Comparisons of Urge to Smoke VAS Parameters Between myblu™ and Continuous Smoking or JUUL Product Following Ad Libitum Use (PK Population) |

## **14.2.6** Questionnaire Tables

## 14.2.6.1 PSCDI or PSECDI Total Score

Table 14.2.6.1.1 Summary of PSCDI or PSECDI Total Score by Study Product and Study Day (ITT Population)

## 14.2.6.2 Cough Questionnaire

Table 14.2.6.2.1 Frequency Count of Cough Questionnaire by Study Product and Study Day (ITT Population)

### 14.2.6.3 MTWS-R Total Score

Table 14.2.6.3.1 Summary of MTWS-R Total Score by Study Product and Study Day (ITT Population)

## 14.2.6.4 **QSU-brief Factor Scores**

Table 14.2.6.4.1 Summary of QSU-brief Factor Scores by Study Product and Study Day (ITT Population)

### 14.2.6.5 PES Subscales

Table 14.2.6.5.1 Summary of PES Subscales by Study Product and Study Day (ITT Population)

## 14.2.6.6 Product Liking VAS Score

Table 14.2.6.6.1 Summary of Product Liking VAS Score by Study Product and Study Day (ITT Population)

### 14.2.6.7 Future Intent to Use VAS Score

Table 14.2.6.7.1 Summary of Future Intent to Use VAS Score by Study Product and Study Day (ITT Population)

## 14.2.6.8 Product and Health Effect Perceptions VAS Score

Table 14.2.6.8.1 Summary of Product and Health Effect Perceptions VAS Score by Study Product and Study Day (ITT Population)

## **14.2.7 Product Use Figures**

| Mean (+/- SD) Self-Reported Number of <i>my</i> blu <sup>™</sup> Pods Started Versus Day (ITT) |
|---|
| Mean Self-Reported Number of <i>my</i> blu <sup>™</sup> Pods Started Versus Day (ITT) |
| Mean (+/- SD) Self-Reported Number of <i>my</i> blu <sup>™</sup> Pods Started Versus Day (PP 28/29) |
| Mean Self-Reported Number of <i>my</i> blu <sup>™</sup> Pods Started Versus Day (PP 28/29) |
| Mean (+/- SD) Self-Reported Number of <i>my</i> blu <sup>TM</sup> Pods Started Versus Day (PP 56/57) |
| Mean Self-Reported Number of <i>my</i> blu <sup>™</sup> Pods Started Versus Day (PP 56/57) |
| Mean (+/- SD) Self-Reported Number of Cigarettes Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (ITT) |
| Mean Self-Reported Number of Cigarettes Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (ITT) |
| Mean (+/- SD) Self-Reported Number of Cigarettes<br>Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (PP 28/29) |
| Mean Self-Reported Number of Cigarettes Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (PP 28/29) |
| Mean (+/- SD) Self-Reported Number of Cigarettes Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (PP 56/57) |
| Mean Self-Reported Number of Cigarettes Smoked Versus Day for <i>my</i> blu <sup>TM</sup> Products (PP 56/57) |

| Figure 14.2.7.13 | Mean (+/- SD) Self-Reported Number of Cigarettes<br>Smoked Versus Day for Subject's Usual Brand<br>Combustible Cigarette (ITT) |
|---|---|
| Figure 14.2.7.14 | Mean Self-Reported Number of Cigarettes Smoked<br>Versus Day for Subject's Usual Brand Combustible<br>Cigarette (ITT) |
| Figure 14.2.7.15 | Mean (+/- SD) Self-Reported Number of Cigarettes<br>Smoked Versus Day for Subject's Usual Brand<br>Combustible Cigarette (PP 28/29) |
| Figure 14.2.7.16 | Mean Self-Reported Number of Cigarettes Smoked<br>Versus Day for Subject's Usual Brand Combustible<br>Cigarette (PP 28/29) |
| Figure 14.2.7.17 | Mean (+/- SD) Self-Reported Number of Cigarettes<br>Smoked Versus Day for Subject's Usual Brand<br>Combustible Cigarette (PP 56/57) |
| Figure 14.2.7.18 | Mean Self-Reported Number of Cigarettes Smoked<br>Versus Day for Subject's Usual Brand Combustible<br>Cigarette (PP 56/57) |

# 14.2.8 Biomarker Figures

## 14.2.8.1 Whole Blood COHb

| Figure 14.2.8.1.1.1 | Arithmetic Mean (SD) Whole Blood COHb by Study<br>Product and Study Day (ITT Population) |
|---|---|
| Figure 14.2.8.1.1.2 | Arithmetic Mean (SD) Whole Blood COHb by Study<br>Product and Study Day (PP Population) |
| Figure 14.2.8.1.2.1 | Arithmetic Mean (SD) Whole Blood COHb Change<br>From Baseline by Study Product and Study Day (ITT<br>Population) |
| Figure 14.2.8.1.2.2 | Arithmetic Mean (SD) Whole Blood COHb Change<br>From Baseline by Study Product and Study Day (PP<br>Population) |
| Figure 14.2.8.1.3.1 | Arithmetic Mean (SD) Whole Blood COHb Percent<br>Change From Baseline by Study Product and Study<br>Day (ITT Population) |
| Figure 14.2.8.1.3.2 | Arithmetic Mean (SD) Whole Blood COHb Percent<br>Change From Baseline by Study Product and Study<br>Day (PP Population) |

## **14.2.8.2** Urine NNAL

Figure 14.2.8.2.1.1 Arithmetic Mean (SD) Urine NNAL Amount Excreted by Study Product and Study Day (ITT Population)

| Figure 14.2.8.2.1.2 | Arithmetic Mean (SD) Urine NNAL Amount Excreted<br>by Study Product and Study Day (PP Population) |
|---|---|
| Figure 14.2.8.2.2.1 | Arithmetic Mean (SD) Urine NNAL Amount Excreted<br>Change From Baseline by Study Product and Study<br>Day (ITT Population) |
| Figure 14.2.8.2.2.2 | Arithmetic Mean (SD) Urine NNAL Amount Excreted<br>Change From Baseline by Study Product and Study<br>Day (PP Population) |
| Figure 14.2.8.2.3.1 | Arithmetic Mean (SD) Urine NNAL Amount Excreted<br>Percent Change From Baseline by Study Product and<br>Study Day (ITT Population) |
| Figure 14.2.8.2.3.2 | Arithmetic Mean (SD) Urine NNAL Amount Excreted<br>Percent Change From Baseline by Study Product and<br>Study Day (PP Population) |
| Figure 14.2.8.2.4.1 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine Creatinine by Study Product and Study Day (ITT Population) |
| Figure 14.2.8.2.4.2 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine Creatinine by Study Product and Study Day (PP Population) |
| Figure 14.2.8.2.5.1 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine<br>Creatinine Change From Baseline by Study Product and<br>Study Day (ITT Population) |
| Figure 14.2.8.2.5.2 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine<br>Creatinine Change From Baseline by Study Product and<br>Study Day (PP Population) |
| Figure 14.2.8.2.6.1 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine<br>Creatinine Percent Change From Baseline by Study<br>Product and Study Day (ITT Population) |
| Figure 14.2.8.2.6.2 | Arithmetic Mean (SD) Urine NNAL Adjusted for Urine<br>Creatinine Percent Change From Baseline by Study<br>Product and Study Day (PP Population) |

## 14.2.8.3 Urine 3-HPMA

Figures 14.2.8.3.1.1 through 14.2.8.3.6.2 will be generated for Urine 3-HPMA similar to Urine NNAL.

## **14.2.8.4 Urine S-PMA**

Figures 14.2.8.4.1.1 through 14.2.8.4.6.2 will be generated for Urine S-PMA similar to Urine NNAL.

### 14.2.8.5 Urine NNN

Figures 14.2.8.5.1.1 through 14.2.8.5.6.1, as applicable (ITT population only) will be generated for Urine NNN similar to Urine NNN.

## **14.2.8.6 Urine CEMA**

Figures 14.2.8.6.1.1 through 14.2.8.6.6.1, as applicable (ITT population only) will be generated for Urine CEMA similar to Urine NNAL.

### **14.2.8.7 Urine HEMA**

Figures 14.2.8.7.1.1 through 14.2.8.7.6.1, as applicable (ITT population only) will be generated for Urine HEMA similar to Urine NNAL.

### **14.2.8.8 Urine HMPMA**

Figures 14.2.8.8.1.1 through 14.2.8.8.6.1, as applicable (ITT population only) will be generated for Urine HMPMA similar to Urine NNAL.

### **14.2.8.9 Urine MHBMA**

Figures 14.2.8.9.1.1 through 14.2.8.9.6.1, as applicable (ITT population only) will be generated for Urine MHBMA similar to Urine NNAL.

### 14.2.8.10 Urine 1-OHP

Figures 14.2.8.10.1.1 through 14.2.8.10.6.1, as applicable (ITT population only) will be generated for Urine 1-OHP similar to Urine NNAL.

### 14.2.8.11 Urine o-tol

Figures 14.2.8.11.1.1 through 14.2.8.11.6.1, as applicable (ITT population only) will be generated for Urine o-tol similar to Urine NNAL.

## 14.2.8.12 Urine 3-OH B[a]P

Figures 14.2.8.12.1.1 through 14.2.8.12.6.1, as applicable (ITT population only) will be generated for Urine 3-OH B[a]P similar to Urine NNAL.

## 14.2.8.13 Urine 1-AN

Figures 14.2.8.13.1.1 through 14.2.8.13.6.1, as applicable (ITT population only) will be generated for Urine 1-AN similar to Urine NNAL.

#### 14.2.8.14 Urine 2-AN

Figures 14.2.8.14.1.1 through 14.2.8.14.6.1, as applicable (ITT population only) will be generated for Urine 2-AN similar to Urine NNAL.

## **14.2.8.15** Urine Nicotine Equivalents

Figures 14.2.8.15.1.1 through 14.2.8.15.6.1, as applicable (ITT population only) will be generated for Urine Nicotine Equivalents similar to Urine NNAL.

### 14.2.8.16 Plasma sICAM

Figures 14.2.8.16.1.1 through 14.2.8.16.31, as applicable (ITT population only) will be generated for Plasma sICAM similar to Whole Blood COHb.

### 14.2.8.17 Whole Blood WBCs

Figures 14.2.8.17.1.1 through 14.2.8.17.3.1, as applicable (ITT population only) will be generated for Whole Blood WBCs similar to Whole Blood COHb.

#### **14.2.8.18 Serum HDL-C**

Figures 14.2.8.18.1.1 through 14.2.8.18.3.1, as applicable (ITT population only) will be generated for Serum HDL-C similar to Whole Blood COHb.

### 14.2.8.19 Serum MCP-1

Figures 14.2.8.19.1.1 through 14.2.8.19.3.1, as applicable (ITT population only) will be generated for Serum MCP-1 similar to Whole Blood COHb.

## 14.2.8.20 Urine Type III isoprostane (8-epi-prostaglandin F2α)

Figures 14.2.8.20.1.1 through 14.2.8.20.6.1, as applicable (ITT population only) will be generated for Urine Type III isoprostane (8-epi-prostaglandin  $F2\alpha$ ) similar to Urine NNAL.

### 14.2.8.21 Urine 11-dehydrothromboxane B2

Figures 14.2.8.21.1.1 through 14.2.8.21.6.1, as applicable (ITT population only) will be generated for Urine 11-dehydrothromboxane B2 similar to Urine NNAL.

## 14.2.9 Physiologic Assessments Figures

#### 14.2.9.1 FeNO

Figures 14.2.8.22.1.1 through 14.2.8.22.3.1, as applicable (ITT population only) will be generated for FeNO similar to Whole Blood COHb.

## 14.2.9.2 Systolic Blood Pressure

Figures 14.2.9.2.1.1 through 14.2.9.2.3.1, as applicable (ITT population only) will be generated for Systolic Blood Pressure similar to Whole Blood COHb.

## 14.2.9.3 Diastolic Blood Pressure

Figures 14.2.9.3.1.1 through 14.2.9.3.3.1, as applicable (ITT population only) will be generated for Diastolic Blood Pressure similar to Whole Blood COHb.

### **14.2.9.4 Heart Rate**

Figures 14.2.9.4.1.1 through 14.2.9.4.3.1, as applicable (ITT population only) will be generated for Heart Rate similar to Whole Blood COHb.

| 14.2.10 P | harmacokinetics Figures |
|---|---|
| Figure 14.2.10.1 | Arithmetic Mean (SD) Unadjusted Plasma Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (PK Population) |
| Figure 14.2.10.2 | Arithmetic Mean Plasma Unadjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (PK Population) |
| Figure 14.2.10.3 | Arithmetic Mean Plasma Unadjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Semi-log Scale) (PK Population) |
| Figure 14.2.10.4 | Arithmetic Mean (SD) Baseline-adjusted Plasma<br>Nicotine Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (PK Population) |
| Figure 14.2.10.5 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Linear Scale) (PK Population) |
| Figure 14.2.10.6 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following<br>Controlled Use (Semi-log Scale) (PK Population) |
| Figure 14.2.10.7 | Arithmetic Mean (SD) Unadjusted Plasma Nicotine<br>Concentration Versus Time Profiles Following Ad<br>Libitum Use (Linear Scale) (PK Population) |
| Figure 14.2.10.8 | Arithmetic Mean Plasma Unadjusted Nicotine<br>Concentration Versus Time Profiles Following Ad<br>Libitum Use (Linear Scale) (PK Population) |

| Figure 14.2.10.9 | Arithmetic Mean Plasma Unadjusted Nicotine<br>Concentration Versus Time Profiles Following Ad<br>Libitum Use (Semi-log Scale) (PK Population) |
|---|---|
| Figure 14.2.10.10 | Arithmetic Mean (SD) Baseline-adjusted Plasma<br>Nicotine Concentration Versus Time Profiles Following<br>Ad Libitum Use (Linear Scale) (PK Population) |
| Figure 14.2.10.11 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following Ad<br>Libitum Use (Linear Scale) (PK Population) |
| Figure 14.2.10.12 | Arithmetic Mean Plasma Baseline-adjusted Nicotine<br>Concentration Versus Time Profiles Following Ad<br>Libitum Use (Semi-log Scale) (PK Population) |

Note: Individual profiles will be presented in an appendix of the report.

## 14.2.11 Urge to Smoke Figures

| Figure 14.2.11.1 | Arithmetic Mean (SD) of Urge to Smoke by Study |
|---|---|
| | Product Following Ad Libitum Use (PK Population) |
| Figure 14.2.11.2 | Arithmetic Mean (SD) of Baseline-adjusted Urge to<br>Smoke by Study Product Following Ad Libitum Use |
| | (PK Population) |

## 14.2.12 Questionnaire Figures

## 14.2.12.1 PSCDI or PSECDI Total Score

Figure 14.2.12.1.1 Box plot of PSCDI or PSECDI Total Score by Study Product and Study Day (ITT Population)

#### 14.2.12.2 MTWS-R Total Score

Figure 14.2.12.2.1 Arithmetic Mean (SD) MTWS-R Total Score by Study Product and Study Day (ITT Population)

### 14.2.12.3 QSU-brief Factor Scores

- Figure 14.2.12.3.1.1 Arithmetic Mean (SD) QSU-brief Factor Scores (Factor 1) by Study Product and Study Day (ITT Population)
- Figure 14.2.12.3.2.1 Arithmetic Mean (SD) QSU-brief Factor Scores (Factor 2) by Study Product and Study Day (ITT Population)

## **14.2.12.4 PES Subscales**

- Figure 14.2.12.4.1.1 Arithmetic Mean (SD) PES Subscales (Satisfaction) by Study Product and Study Day (ITT Population)
- Figure 14.2.12.4.2.1 Arithmetic Mean (SD) PES Subscales (Psychological Reward) by Study Product and Study Day (ITT Population)

| Figure 14.2.12.4.3.1 | Arithmetic Mean (SD) PES Subscales (Aversion) by<br>Study Product and Study Day (ITT Population) |
|---|---|
| Figure 14.2.12.4.4.1 | Arithmetic Mean (SD) PES Subscales (Relief) by Study<br>Product and Study Day (ITT Population) |
| Figure 14.2.12.4.5.1 | Arithmetic Mean (SD) PES Subscales (Item 17) by<br>Study Product and Study Day (ITT Population) |
| Figure 14.2.12.4.6.1 | Arithmetic Mean (SD) PES Subscales (Item 19) by<br>Study Product and Study Day (ITT Population) |
| Figure 14.2.12.4.7.1 | Arithmetic Mean (SD) PES Subscales (Item 21) by<br>Study Product and Study Day (ITT Population) |

### 14.2.12.5 Product Liking VAS Score

Figure 14.2.12.5.1 Arithmetic Mean (SD) Product Liking VAS Score by Study Product and Study Day (ITT Population)

#### 14.2.12.6 Future Intent to Use VAS Score

Figure 14.2.12.6.1 Arithmetic Mean (SD) Future Intent to Use VAS Score by Study Product and Study Day (ITT Population)

## 14.2.12.7 Product and Health Effect Perceptions VAS Score

- Figure 14.2.12.7.1.1 Arithmetic Mean (SD) Product and Health Effect
  Perceptions VAS Score (Question 1) by Study Product
  and Study Day (ITT Population)
- Figure 14.2.12.7.2.1 Arithmetic Mean (SD) Product and Health Effect
  Perceptions VAS Score (Question 2) by Study Product
  and Study Day (ITT Population)
- Figure 14.2.12.7.3.1 Arithmetic Mean (SD) Product and Health Effect
  Perceptions VAS Score (Question 3) by Study Product
  and Study Day (ITT Population)
- Figure 14.2.12.7.4.1 Arithmetic Mean (SD) Product and Health Effect Perceptions VAS Score (Question 4) by Study Product and Study Day (ITT Population)

## 14.3 Safety Data Summary Tables

### 14.3.1 Displays of Adverse Events

Table 14.3.1.1 Product Use-emergent Adverse Event Frequency by Study Product – Number of Subjects Reporting the Event (% of Subjects Who Used Study Product) (Safety Population)

- Table 14.3.1.2 Product Use-emergent Adverse Event Frequency by Study Product Number of Adverse Events (% of Total Adverse Events) (Safety Population)
- Table 14.3.1.3 Product Use-emergent Adverse Event Frequency by Study Product, Severity, and Relationship to Study Product Number of Subjects Reporting Events (Safety Population)

## 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population) <if no serious adverse event occurred, a statement 'No serious adverse event is reported'>

# 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

### 14.3.4 Abnormal Laboratory Value Listing (each subject)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology (Safety Population)
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis (Safety Population)
- Table 14.3.4.4 Clinically Significant Values and Recheck Results (Safety Population)

# 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary Serum Chemistry (Safety Population)
- Table 14.3.5.2 Clinical Laboratory Summary Hematology (Safety Population)
- Table 14.3.5.3 Clinical Laboratory Summary Urinalysis (Safety Population)
- Table 14.3.5.4 Vital Sign Summary (Safety Population)
- Table 14.3.5.5 12-Lead Electrocardiogram Summary (Safety Population)
- Table 14.3.5.6 Spirometry Summary (Safety Population)

### **Section 16 Data Listings**

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

## **16.1** Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

## 16.2 Subject Data Listings

## **16.2.1** Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (Safety Population)

### **16.2.2 Protocol Deviations**

Appendix 16.2.2 Protocol Deviations

## 16.2.3 Subjects Excluded from Analysis

Appendix 16.2.3 Subjects Excluded from Analysis

Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the study report.

## 16.2.4 Demographic Data

| Appendix 16.2.4.1.1 | Subject Information (Safety Population) |
|---------------------|-----------------------------------------|
| Appendix 16.2.4.1.2 | Demographics (Safety Population) |

Appendix 16.2.4.1.3 Additional Demographics Questionnaire (Safety Population)

Appendix 16.2.4.2.1 Physical Examination – Full (Safety Population)

Appendix 16.2.4.2.2 Physical Examination - Symptom-driven (Safety Population)

Appendix 16.2.4.3 Medical and Surgical History (Safety Population)

Appendix 16.2.4.4.1 Tobacco/Nicotine Product Use History Questionnaire (Safety Population)

Appendix 16.2.4.4.2 Smoking History (Safety Population)

Appendix 16.2.4.4.3 Usual Brand Documentation (Safety Population)

## 16.2.5 Compliance and/or Concentration Data

Appendix 16.2.5.1 Inclusion / Exclusion Criteria Not Met (Safety Population)

# Clinical Study Report No. CA22747

| <br>icai Study Report No. | |
|---|---|
| Appendix 16.2.5.2.1 | <i>my</i> blu <sup>TM</sup> Product Preference Questionnaire (Safety Population) |
| Appendix 16.2.5.2.2 | Product Selection (Safety Population) |
| Appendix 16.2.5.2.3 | Staff-Recorded In-Clinic Product Use (Safety Population) |
| Appendix 16.2.5.2.4 | Self-Reported Product Use (Safety Population) |
| Appendix 16.2.5.2.5 | Product Use - Nicotine PK Assessment (Safety Population) |
| Appendix 16.2.5.3.1 | Pharmacokinetics Blood Sampling (Safety Population) |
| Appendix 16.2.5.3.2 | 24-Hour Urine Collection (Safety Population) |
| Appendix 16.2.5.3.3 | 24-Hour Urine Collection - Pod Weight Documentation (Safety Population) |
| Appendix 16.2.5.3.4 | Carboxyhemoglobin Blood Collection (Safety Population) |
| Appendix 16.2.5.3.5 | Biomarkers and Bio-Banking Blood Collection (Safety Population) |
| Appendix 16.2.5.4 | Concomitant Medications (Safety Population) |
| 16.2.6 | Individual, Biomarker, Pharmacokinetics and |
| | Subjective Effect Data |
| Appendix 16.2.6.2.1 | Whole Blood COHb* |
| Appendix 16.2.6.2.1<br>Appendix 16.2.6.2.2 | Whole Blood COHb* |
| 11 | Whole Blood COHb* Urine NNAL* |
| Appendix 16.2.6.2.2 | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* |
| Appendix 16.2.6.2.2<br>Appendix 16.2.6.2.3<br>Appendix 16.2.6.2.4 | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* nclude population flags in these listings to show who |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* nclude population flags in these listings to show who |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* Include population flags in these listings to show who opulation. |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* Include population flags in these listings to show who epulation. Urine NNN (ITT Population) |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po Appendix 16.2.6.2.5 Appendix 16.2.6.2.6 Appendix 16.2.6.2.7 | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* Include population flags in these listings to show who opulation. Urine NNN (ITT Population) Urine CEMA (ITT Population) |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po Appendix 16.2.6.2.5 Appendix 16.2.6.2.6 Appendix 16.2.6.2.7 Appendix 16.2.6.2.8 | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* Include population flags in these listings to show who equivariantly appropriate to the second |
| Appendix 16.2.6.2.2 Appendix 16.2.6.2.3 Appendix 16.2.6.2.4 * Programmer note: I was in ITT and PP po Appendix 16.2.6.2.5 Appendix 16.2.6.2.6 Appendix 16.2.6.2.7 Appendix 16.2.6.2.8 Appendix 16.2.6.2.9 | Whole Blood COHb* Urine NNAL* Urine 3-HPMA* Urine S-PMA* Include population flags in these listings to show who opulation. Urine NNN (ITT Population) Urine CEMA (ITT Population) Urine HEMA (ITT Population) Urine HMPMA (ITT Population) |

Appendix 16.2.6.2.11 Urine o-tol (ITT Population)

Appendix 16.2.6.2.12 Urine 3-OH B[a]P (ITT Population) Appendix 16.2.6.2.13 Urine 1-AN (ITT Population) Appendix 16.2.6.2.14 Urine 2-AN (ITT Population) Appendix 16.2.6.2.15.1 Urine Nicotine and Metabolites (ITT Population) Appendix 16.2.6.2.15.2 Urine Nicotine Equivalents (ITT Population) Appendix 16.2.6.2.16 Plasma sICAM (ITT Population) Appendix 16.2.6.2.17 Whole Blood WBCs (ITT Population) Appendix 16.2.6.2.18 Serum HDL-C (ITT Population) Appendix 16.2.6.2.19 Serum MCP-1 (ITT Population) Appendix 16.2.6.2.20 Urine Type III isoprostane (8-epi-prostaglandin  $F2\alpha$ ) (ITT Population) Appendix 16.2.6.2.21 Urine 11-dehydrothromboxane B2 (ITT Population) Appendix 16.2.6.3.1 PSCDI, PSECDI Questionnaire (ITT Population) Appendix 16.2.6.3.2 PSCDI, PSECDI Questionnaire Responses (ITT **Population** Appendix 16.2.6.4.1 Cough Questionnaire (ITT Population) Appendix 16.2.6.4.2 Cough Questionnaire Responses (ITT Population) Appendix 16.2.6.5.1 MTWS-R Questionnaire (ITT Population) Appendix 16.2.6.5.2 MTWS-R Questionnaire Responses (ITT Population) Appendix 16.2.6.6.1 QSU-brief Questionnaire (ITT Population)

- Appendix 16.2.6.7.1 PES Questionnaire (ITT Population)
- Appendix 16.2.6.7.2 PES Questionnaire Responses (ITT Population)

Appendix 16.2.6.6.2 QSU-brief Questionnaire Responses (ITT Population)

- Appendix 16.2.6.7.3 PES Questionnaire Subscales (ITT Population)
- Appendix 16.2.6.8 Product Liking Questionnaire Responses (ITT Population)

| nical Study Report No. | CA22747 |
|---|---|
| Appendix 16.2.6.9 | Future Intent to Use Questionnaire Responses (ITT Population) |
| Appendix 16.2.6.10 | Product and Health Effect Perceptions Questionnaire<br>Responses (ITT Population) |
| 16.2.7 Adverse Ev | ents Listings |
| Appendix 16.2.7.1.1 | Adverse Events (I of II) (Safety Population) |
| Appendix 16.2.7.1.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.2 | Adverse Event Non- Medication Therapy (Safety Population) |
| Appendix 16.2.7.3 | Adverse Event Preferred Term Classification (Safety Population) |
| 16.2.8 Listings of Safety Obse | Individual Laboratory Measurements and Other ervations |
| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety |
| | Population) |
| Appendix 16.2.8.1.2 | • • |
| Appendix 16.2.8.1.2 Appendix 16.2.8.1.3 | Population) Clinical Laboratory Report - Hematology (Safety |
| | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety |
| Appendix 16.2.8.1.3 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 Appendix 16.2.8.1.5 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) Urine Drug Screen (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 Appendix 16.2.8.1.5 Appendix 16.2.8.1.6 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) Urine Drug Screen (Safety Population) Alcohol Breath Test (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 Appendix 16.2.8.1.5 Appendix 16.2.8.1.6 Appendix 16.2.8.1.7 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) Urine Drug Screen (Safety Population) Alcohol Breath Test (Safety Population) Urine Cotinine Screen (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 Appendix 16.2.8.1.5 Appendix 16.2.8.1.6 Appendix 16.2.8.1.7 Appendix 16.2.8.1.8 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) Urine Drug Screen (Safety Population) Alcohol Breath Test (Safety Population) Urine Cotinine Screen (Safety Population) Pregnancy Test (Safety Population) |
| Appendix 16.2.8.1.3 Appendix 16.2.8.1.4 Appendix 16.2.8.1.5 Appendix 16.2.8.1.6 Appendix 16.2.8.1.7 Appendix 16.2.8.1.8 Appendix 16.2.8.1.9 | Population) Clinical Laboratory Report - Hematology (Safety Population) Clinical Laboratory Report - Urinalysis (Safety Population) Serology (Safety Population) Urine Drug Screen (Safety Population) Alcohol Breath Test (Safety Population) Urine Cotinine Screen (Safety Population) Pregnancy Test (Safety Population) Serum FSH (Safety Population) |

## 10. TABLE AND FIGURE SHELLS

Appendix 16.2.8.5 Appendix 16.2.8.6

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be presented and included in the final report. Unless otherwise

FeNO Measurement (Safety Population)

Spirometry (Safety Population)

| Nerudia Ltd. |
|-----------------------------------|
| nyblu E-cigarettes |
| Clinical Study Report No. CA22747 |

noted, all tables will be presented in Times New Roman font size 8. These tables will be generated off of the ADaM Version 1.0.

## 10.1 Figures Shells

In-text and post-text PK Figures of mean plasma concentrations and UTS on linear scale will be in the following format: Figure 11-X, 14.X, and appendix 16.2.6.1:

Figure X.X: Arithmetic Mean Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following <Controlled or Ad Libitum> Product Use by Product (Linear Scale) (PK Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

### Notes for Generating the Actual Mean Figure:

- I. Legend will be the short description
- II. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for PK figures and "Urge to Smoke" for UTS figure
- III. X axis label will be "Minutes from Product Use" for all figures

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam meangraph.sas DDMMYYYY HH:MM

Post-text PK Figures of mean (SD) plasma concentrations and UTS on linear scale will be in the following format: Figure 14.X:

Figure 14.X: Arithmetic Mean (SD) Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following < Controlled or Ad Libitum > Product Use by Product (Linear Scale) (PK Population)



Treatments B and C are shifted to the right for ease of reading

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

# Nerudia Ltd. *my*blu E-cigarettes

## Clinical Study Report No. CA22747

## Notes for Generating the Actual Mean Figure:

- IV. Legend will be the short description
- V. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for PK figures and "Urge to Smoke" for UTS figure
  VI. X axis label will be "Minutes from Product Use" for all figures
- VII. Please add the footnote for products that are shifted to the right for ease of reading

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYYY HH:MM Post-text PK Figures of mean plasma concentrations on semi-log scale will be in the following format: 14.X, and appendix 16.2.6.1:

Figure 14.X: Arithmetic Mean Baseline-Adjusted Plasma Nicotine Concentration-Time Profiles Following <Controlled or Ad Libitum> Product Use by Product (Semi-Log Scale) (PK Population)



## Notes for Generating the Actual Mean Figure:

VIII. Legend will be the short descriptions

IX. Y axis label will be "Plasma Nicotine Concentration (ng/mL)" for all figures

X. X axis label will be "Minutes from Product Use" for all figures

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam meangraph.sas DDMMYYYY HH:MM

Clinical Study Report No. CA22747

Post-text Figure(s) for Total Scores will be in the following format:

Figure 14.X: Box Plot of PSCDI or PSECDI Total Score by Study Product and Study Day (ITT Population)

\*\*\*Please note this will be a boxplot figure\*\*\*

### Notes for Generating the Actual Mean Figure:

- XI. Note: this figure will be a boxplot figure
- XII. Please present each subjective measurement on different graphs but associated with Figure 14.2.9.1 or similar graphs. Present each question (or factor scale, subscale, or total score) in the title of each graph.
- XIII. Y axis label will be "Subjective Measurement Score"
- XIV. X axis label will be labelled with "A, B, C, D, E, F" for each figure representing each product

# 10.2 Post-Text Summary Tables Shells

## 14.1 Demographic Tables

Table 14.1.1 Summary of Disposition (Safety, ITT, and PP Populations)

| | | | P: | roduct | | | | |
|------------|--------------------|----|----|--------|----|----|----|---------|
| Population | Category | Α | В | С | D | E | F | Overall |
| Safety | Enrolled | | | | | | | XX |
| | Randomized | XX | XX | XX | XX | XX | XX | XX |
| | Completed | XX | XX | XX | XX | XX | XX | XX |
| | Discontinued Early | X | X | X | X | X | X | X |
| | <reason></reason> | X | X | X | X | X | Χ | X |
| ITT | Enrolled | | | | | | | XX |
| | Randomized | XX | XX | XX | XX | XX | XX | XX |
| | Completed | XX | XX | XX | XX | XX | XX | XX |
| | Discontinued Early | X | X | X | X | X | X | X |
| | <reason></reason> | X | X | X | Χ | X | Χ | X |
| PP | Enrolled | | | | | | | XX |
| | Randomized | XX | XX | XX | XX | XX | XX | XX |
| | Completed | XX | XX | XX | XX | XX | XX | XX |
| | Discontinued Early | X | X | X | X | X | X | X |
| | <reason></reason> | X | X | X | X | X | X | X |

Note: Product X: < >

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab prog\_name.sas DDMMMYYYY HH:MM


# Nerudia Ltd. *my*blu E-cigarettes

# Clinical Study Report No. CA22747


Table 14.1.2 Demographic Summary (Safety, ITT, and PP Populations)

| | | | | | | | | Product | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Population | Trait | | | А | | В | | С | | D | | E | | F | 0 | verall |
| Safety | Sex | Male | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X% | Х | (XX.X%)) | X | (XX.X%) |
| | | Female | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X% | Χ | (XX.X%)) | Χ | (XX.X%) |
| | Race | American Indian | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X%) | Х | (XX.X% | Х | (XX.X%)) | Х | (XX.X%) |
| | | Asian | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X% | X | (XX.X%)) | Χ | (XX.X%) |
| | | Black | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X%) | Χ | (XX.X% | Χ | (XX.X%)) | Χ | (XX.X%) |
| | Age(yrs) | n | | X | | X | | X | | X | | X | | X | | X |
| | | Mean | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X |
| | | SD | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX |
| | | Minimum | | XX | | XX | | XX | | XX | | XX | | XX | | XX |
| | | Median | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X |
| | | Maximum | | XX | | XX | | XX | | XX | | XX | | XX | | XX |
| | Weight(kg) | n | | X | | X | | X | | X | | Х | | X | | Х |
| | | Mean | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X |
| | | SD | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX | | X.XX |
| | | Minimum | | XX | | XX | | XX | | XX | | XX | | XX | | XX |
| | | Median | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X | | X.X |
| | | Maximum | | XX | | XX | | XX | | XX | | XX | | XX | | XX |

<Continued with other measures - Body Mass Index  $(kg/m^2)$  and ITT and PP populations.>

Note: Product X: < >

Age is derived from birth date to date of informed consent.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

# Nerudia Ltd. *my*blu E-cigarettes

# Clinical Study Report No. CA22747


Table 14.1.3 Smoking History Summary (Safety, ITT, and PP Populations)

| | | | | | Product | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Population | on Trait | _ | А | В | C | D | E | <br>F | Overall |
| Safety | CPD | n | Х | Х | X | Х | Х | X | Х |
| | | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX | XX |
| | Number of | n | X | Х | X | Х | X | X | X |
| | Years Smoked | Mean | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX | XX |
| | Usual Brand | Menthol | X(XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | Cigarette Flavor | Regular | X (XX%) | X(XX%) | X (XX%) | X (XX%) | X (XX%) | X(XX%) | X (XX%) |

<Continued with ITT and PP populations.>

Note: Product X: < >

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

## Nerudia Ltd.

## *my*blu E-cigarettes

# Clinical Study Report No. CA22747

#### 14.2.1 Main Study Product Use Tables

Note: Product Use (In-Clinic) Tables will have the following format:


Table 14.2.1.1 Summary of In-Clinic Number of myblu™ Pods Started by Product and Day (ITT)

| | | | | Da | У | | |
|------|------|-----------|------|--------|------|------|------|
| Prod | duct | Statistic | -2 | <br>-1 | 1 | 2 | etc. |
| | A | n | X | X | X | X | |
| | | Mean | X.X | X.X | X.X | X.X | |
| | | SD | X.XX | X.XX | X.XX | X.XX | |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X | |
| | | SEM | X.XX | X.XX | X.XX | X.XX | |
| | | Minimum | XX | XX | XX | XX | |
| | | Median | X.X | X.X | X.X | X.X | |
| | | Maximum | XX | XX | XX | XX | |

\_\_\_\_\_\_

Note: Product X: < >

NA: Not applicable

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: Days 1 through 3, 28, 29, 56, and 57 will be presented in Tables 14.2.1.1 through 14.2.1.3. Product E will not be presented in Tables 14.2.1.1 through 14.2.1.6. Only Days 3, 28, 29, 56, and 57 will be presented in Tables 14.2.1.4 through 14.2.1.6. Days -2 through 3 (Days 2 and 3 will be NA for the combustible cigarette group), 28, 29, 56, and 57 will be presented in Tables 14.2.1.7 through 14.2.1.9.

# Nerudia Ltd. *my*blu E-cigarettes

# Clinical Study Report No. CA22747

Note: Product Use (Self-Reported) Tables will have the following format:


Table 14.2.1.10 Summary of Self-Reported Number of myblu™ Pods Started by Product and Day (ITT)

| | | | | ·Day | |
|---------|-----------|------|------|------|------|
| Product | Statistic | 3 | 4 | 5 | 6 |
| A | n | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |
| В | n | X | X | X | Х |
| | Mean | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX |

Note: Product X: < >

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programmer Note: Days 3 through 57 and Products C and D will be presented. Product E also be presented in Tables 14.2.1.16 through 14.2.1.18. Frequency counts (n,%) will be presented as the statistics in Tables 14.2.1.13 through 14.2.1.15.

# Nerudia Ltd. *my*blu E-cigarettes

Clinical Study Report No. CA22747

Note: Summary Tables 14.2.1.19 through 14.2.1.21 will have the following format:

Table 14.2.1.19 Summary of Self-Reported Product Use by Product and Product Use Period (ITT)

| | | | | Pro | oduct | |
|---|---|---|---|---|---|---|
| Variable | Product Use Period | Statistic | А | В | С | D |
| Number of Cigarettes | 1 | n | X | X | X | X |
| _ | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |
| | 2 | n | X | X | X | Х |
| | | Mean | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX |

Note: Product X: < >

NA: Not applicable

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programmer Note: Other variables presented will be Number of myblu<sup>TM</sup> started and >=50 Puffs Taken From myblu<sup>TM</sup>. Frequency counts (n, %) will be presented for >= 50 Puffs Taken From myblu<sup>TM</sup>. Product E will also be presented (NA for all variables except number of cigarettes)


Clinical Study Report No. CA22747

## **14.2 Biomarker Tables**

Tables 14.2.2.1.1.1, 14.2.2.1.1.2, 14.2.2.1.1.3 and other summary tables for ITT population will be in the following format:


Table 14.2.2.1.1.1 Summary of Whole Blood COHb by Study Product and Study Day (ITT Population)

| | | | | Product | | | |
|-------|-----------|------|------|---------|------|------|------|
| Day | Statistic | Α | В | С | D | E | F |
| XXXXX | n | X | X | X | X | X | Х |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |

Note: Product X: < >

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Notes: Footnotes to include under the table, as appropriate: < . = Value missing or not reportable. > The Days will be Day -2 (for some endpoints this may be Day -1), Day 28, and Day 56. For Change from baseline and percent change from baseline, Day -2 will not be presented in the table.

A table should also be presented for PK population for the following biomarkers: NNAL, NNN, 3-HPMA, CEMA, HMPMA, S-PMA; this table shall include Day 3.

Tables 14.2.2.1.1.4, 14.2.2.1.1.5, 14.2.2.1.1.6 and other summary tables for PP population (only for primary biomarkers) will be in the following format:


Table 14.2.2.1.1.4 Summary of Whole Blood COHb by Study Product and Study Day (PP Populations)

| | | PP 2 | 8/29 | PP 56, | /57 | |
|---------|-----------|----------|--------|----------|--------|--------|
| Product | Statistic | Baseline | Day 28 | Baseline | Day 28 | Day 56 |
| A | n | X | X | X | Х | X |
| | Mean | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | CV (%) | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SEM | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX |

\_\_\_\_\_\_

Note: Product X: < >

Program: /CAXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Notes: Footnotes to include under the table, as appropriate: <. = Value missing or not reportable. > Products B through E will also be presented in the table. For Change from baseline and percent change from baseline, Baseline timepoint will not be presented in the table.

# Nerudia Ltd. *my*blu E-cigarettes

Clinical Study Report No. CA22747

## Statistical comparison tables will be in the following format:


Table 14.2.2.1.2.1 Statistical Comparison of Whole Blood COHb Change From Baseline Between myblu™ and Continuous Smoking by Study Day (ITT Population)

| Day | Comparison | Test (n) | S Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| 28 | Product A vs Product E Product B vs Product E Product C vs Product E Product D vs Product E | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |
| 56 | Product A vs Product E<br>Product B vs Product E<br>Product C vs Product E<br>Product D vs Product E | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |

Note: Test = First product in the comparison; Reference = Product E

n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the model.

Product X: < >

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

A table should also be presented for PK population for the following biomarkers: NNAL, NNN, 3-HPMA, CEMA, HMPMA, S-PMA; this table shall include Day 3.

# Nerudia Ltd. *my*blu E-cigarettes

## Clinical Study Report No. CA22747

Table 14.2.2.1.2.2 Statistical Comparison of Whole Blood COHb Change From Baseline Between myblu™ and Continuous Smoking by Study Day (PP Population)

| Day | Comparison | Test (n) | S Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| 28 | Product A vs Product E Product B vs Product E Product C vs Product E Product D vs Product E | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |
| 56 | Product A vs Product E Product B vs Product E Product C vs Product E Product D vs Product E | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |

Note: Test = First product in the comparison; Reference = Product E

n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the model.

Day 28 results are from the Day 28/29 PP Population Day 56 results are from the Day 56/57 PP Population

Product X: < >

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

## Nerudia Ltd.

## *my*blu E-cigarettes

## Clinical Study Report No. CA22747

Statistical Tables 14.2.2.1.3.1 (ITT) and 14.2.2.1.3.2 (PP) will be in the following format:

Table 14.2.2.1.3.1 Statistical Comparison of Whole Blood COHb Change From Baseline Between Day 28 and Day 56 in the myblu™ Groups (ITT Population)

| Product | LS M<br>Day 28 (n) | eans<br>Day 56 (n) | LS Mean Difference<br>(Day 28 - Day 56) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|
| A | X.XX (X) | X.XX (X) | XXX.XX | xx.xx - xxx.xx | X.XXXX |
| В | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| С | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |
| D | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXXX |

Note: n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the model.

Product X: < >

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

## Nerudia Ltd.

# myblu E-cigarettes

## Clinical Study Report No. CA22747

Statistical Table 14.2.2.1.4.1 (ITT) will be in the following format:

Table 14.2.2.1.4.1 Statistical Comparison of Whole Blood COHb Change From Baseline Between myblu™ Groups by Study Day (ITT Population)

| Day | Comparison | Test (n) | S Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| 28 | Product A vs Product B Product A vs Product C Product A vs Product D Product B vs Product C Product B vs Product D Product C vs Product D | X.XX (X) X.XX (X) X.XX (X) X.XX (X) X.XX (X) X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |
| 56 | Product A vs Product B Product A vs Product C Product A vs Product D Product B vs Product C Product B vs Product D Product C vs Product D | X.XX (X) X.XX (X) X.XX (X) X.XX (X) X.XX (X) X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |

Note: Test = First product in the comparison; Reference = Second product in the comparison

n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the model.

Product X: < >

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMYYYYY HH:MM
#### Clinical Study Report No. CA22747

Statistical Table 14.2.2.1.4.2 (PP) will be in the following format:

Table 14.2.2.1.4.2 Statistical Comparison of Whole Blood COHb Change From Baseline Between myblu™ Groups by Study Day (PP Population)

| Day | Comparison | Test (n) | Means<br>Reference (n) | LS Mean Difference<br>(Test - Reference) | 95% Confidence Interval | p-value |
|---|---|---|---|---|---|---|
| 28 | Product A vs Product B Product A vs Product C Product A vs Product D Product B vs Product C Product B vs Product D Product C vs Product D | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |
| 56 | Product A vs Product B Product A vs Product C Product A vs Product D Product B vs Product C Product B vs Product D Product C vs Product D | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X)<br>X.XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX<br>X.XXXX |

Note: Test = First product in the comparison; Reference = Second product in the comparison n = Number of observation used in the analysis; Least-squares means (LS Means) are calculated from the model.

Day 28 results are from the Day 28/29 PP Population Day 56 results are from the Day 56/57 PP Population Product X: < >

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Clinical Study Report No. CA22747

14.2.3 Physiologic Assessments Tables
Physiologic assessments tables (ITT population only), will be similar to Whole Blood COHb (blood biomarker) tables.

Clinical Study Report No. CA22747

#### 14.2.4 Pharmacokinetic Tables and 14.2.5 Urge to Smoke Tables

Tables 14.2.4.1.1.1 through 14.2.4.1.6.2 for unadjusted and Tables 14.2.4.2.1.1 through 14.2.4.2.6.2 for baseline-adjusted concentration data and Tables 14.2.5.1 through 14.2.5.6 for UTS data will be in the following format:

Table 14.2.4.1.1.1 Unadjusted Plasma Nicotine Concentrations (ng/mL) Following Controlled Use of myblu™ closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 2.5 % (Product A) (PK Population)

| Subject | Product Use | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Sequence | Product | Pre-use | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | XXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | | • | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as 1/2 LLOQ. . = Value missing or not reportable.

#### Nerudia Ltd.

#### myblu E-cigarettes

Clinical Study Report No. CA22747

#### Notes for Generating the Actual Table:

Presentation of Data:

For baseline-adjusted table, Pre-use will be replaced with 0.

Concentrations will be presented to same precision as in bio data.

Summary statistics presentation with respect to the precision of the bio data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

Programmer Note:

PK Time points are: pre-use and 3, 5, 7, 10, 12, 15, 20, 30, 60, 120 and 180 minutes following the start of each product use (Controlled and ad libitum)

Please also present the geometric mean and 95% CI around the geometric mean for all concentration tables

Delete the Product Use Sequence column and Product Column as not applicable for parallel studies

Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_conc.sas DDMMYYYY HH:MM

### Tables 14.2.4.3.1.1 through 14.2.4.3.6.2 (PK) and Tables 14.2.5.7 through 14.2.5.12 (UTS) will be in the following format:

Table 14.2.4.3.1.1: Baseline Adjusted Plasma Nicotine Pharmacokinetic Parameters Following Controlled Use of myblu™ Closed System With CF Cosmic Fog Chilled Tobacco Flavor (25 mg With Lactic Acid) (Product A) (PK Population)

| param(<br>(units) | | | param3<br>(units) | | paraml<br>(units) | Product | Product Use<br>Sequence | Subject<br>Number |
|---|---|---|---|---|---|---|---|---|
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | X.XX | X | XXX | X |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | X |
| XX | XX | XX | XX | XX | XX | | | n |
| X.XXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Mean |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SD |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | CV% |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SEM |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | | | Minimum |
| X.XXX | XX.XX | XXX.X | XXX.X | X.XXX | XX.XX | | | Median |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | | | Maximum |
| X.XXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Geom Mean |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | Geom CV% |

<sup>. =</sup> Value missing or not reportable.

Clinical Study Report No. CA22747

#### Notes for Generating the Actual Table:

#### Presentation of Data:

- PK Parameters will be presented in the following order and with following units: AUCO-t (ng\*min/mL), Cmax (ng/mL), Tmax (min)
- n will be presented as an integer (with no decimal);
- Parameter values for exposure based parameters (i.e. AUCO-t and Cmax) will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received). Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean+1; SD and SEM +2, Min and Max +0.
- Values for time-based parameters (i.e. Tmax) will be presented with 2 decimals. Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD +2, Min and Max +0.
- CV% and Geom CV% for all parameters will be presented with 1 decimal
- Delete the Product Use Sequence column and Product Column as not applicable for parallel studies.

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMYYYY HH:MM

#### Tables 14.2.4.4.1.1 and 14.2.4.4.1.2 (PK) and Table 14.2.5.13 (UTS) will be in the following format:

Table 14.2.4.4.1.1: Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameters AUCO-t and Cmax Between myblu™
Products and Continuous Smoking or JUUL Following Controlled Use (PK Population)

| Comparison | Parameter | | etric<br>Means<br>Reference (n) | | Confidence Intervals<br>(95% Confidence) | p-value |
|---|---|---|---|---|---|---|
| Product A vs Product E | AUCO-t<br>Cmax | | X.XX (X)<br>X.XX (X) | | XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXX<br>X.XXX |
| Product B vs Product E | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product C vs Product E | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product D vs Product E | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product A vs Product F | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product B vs Product F | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product C vs Product F | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| Product D vs Product F | AUCO-t | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |
| | Cmax | X.XX (X) | X.XX (X) | XXX.XX | XX.XX - XXX.XX | X.XXX |

Test = The first product in the comparison; Reference = The second product in the comparison n = Number of observations used in the analysis

Product A = myblu™ closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 2.5 % Product B = myblu™ closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 4.0% Product C = myblu™ closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 2.5 % Product D = myblu™ closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 4.0% Product E = Subject's usual brand combustible cigarette

Product F = JUUL® system with Virginia Tobacco Flavor JUULpod, 5.0% nicotine

The mixed model includes product arm, study day, and product arm by study day interaction as fixed effect and subject as a random effect. Parameters are log-transformed prior to analysis. Geometric least-squares means (LS Means) are calculated by exponentiating the LS Means from the ANOVA.

% Geometric LS Mean Ratio = 100\*(Test Product/Reference Product)
Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Tables 14.2.4.4.2.1 and 14.2.4.4.2.2 will be in the following format:

Table 14.2.4.4.2.1: Nonparametric Statistical Comparisons of Baseline-Adjusted Plasma Nicotine PK Parameter Tmax Between myblu™ and Continuous Smoking or JUUL Following Controlled Use (PK Population)

| Comparison | -<br>Parameter | Pro<br>Test | oduct<br>Reference | Differen<br>95% CI | ce Test-Ref<br>Median | erence<br>p-Value |
|---|---|---|---|---|---|---|
| Product A vs Product E | Tmax | X.XX | X.XX | X.XX - X.XX | X.XX | X.XXXX |
| Product B vs Product E | Tmax | X.XX | X.XX | X.XX - X.XX | X.XX | X.XXXX |
| Product C vs Product E | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXXX |
| Product D vs Product E | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXXX |
| Product A vs Product F | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXXX |
| Product B vs Product F | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXXX |
| Product C vs Product F | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXXX |
| Product D vs Product F | Tmax | X.XX | X.XX | x.xx - x.xx | X.XX | X.XXX |

Test = The first product in the comparison; Reference = The second product in the comparison

```
Product A = myblu<sup>m</sup> closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 2.5 % Product B = myblu<sup>m</sup> closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 4.0% Product C = myblu<sup>m</sup> closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 2.5 % Product D = myblu<sup>m</sup> closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 4.0% Product E = Subject's usual brand combustible cigarette Product F = JUUL® system with Virginia Tobacco Flavor JUUL pod, 5.0% nicotine
```

p-values are from Wilcoxon rank sum test.

Program: /CAXXXXX/ECR/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### **14.2.6 Questionnaires Tables**

Tables 14.2.6.1.1-2, 14.2.6.3.1-2, 14.2.6.4.1-2, 14.2.6.5.1-2, 14.2.6.5.1-2, 14.2.6.7.1-2, and 14.2.6.8.1-2 will be in the following format:

Table 14.2.6.1.1 Summary of PSCDI or PSECDI Total Score by Study Product and Study Visit (ITT Population)

| | | Product | | | | | |
|---|---|---|---|---|---|---|---|
| Study Visit | Statistic | A | В | С | D | E | F |
| XXXXXXXX | n | Х | Х | Х | Х | Х | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | Х.Х |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |
| XXXXXXX | n | Х | X | X | X | X | X |
| | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX | XX | XX |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | Maximum | XX | XX | XX | XX | XX | XX |

\_\_\_\_\_\_

Product A =  $myblu^{\text{TM}}$  closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 2.5 % Product B =  $myblu^{\text{TM}}$  closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 4.0%

Product  $C = myblu^m$  closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 2.5 %

Product D = myblu™ closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 4.0%

Product E = Subject's usual brand combustible cigarette

Total scoring: 0 - 3 = not dependent, 4 - 8 = low dependence, 9 - 12 = medium dependence, 13+ = high dependence

Program: /AAXXXXX/ECR/sas prg/stsas/tab programname.sas DDMMMYYYY HH:MM

Programmer note: A table should also be presented for PK population; this table shall include Day 3

Clinical Study Report No. CA22747

Programmer note: When there are multiple scores in a questionnaire to be summarized, an additional column for score category will be added to the table.

#### Nerudia Ltd.

#### myblu E-cigarettes

Clinical Study Report No. CA22747

#### Tables 14.2.6.2.1-2 will be in the following format:

Table 14.2.6.1.1 Frequency Count of Cough Questionnaire by Study Product and Study Visit (ITT Population)

| | | | Product | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | Question | Response | | А | E | 3 | | : | | D | Е | <br>C | | F |
| XXXXXXXX | XXXXXXX | XXXX<br>XXXX<br>XXXX | Χ | (X%)<br>(X%)<br>(X%) | | (X%)<br>(X%)<br>(X%) | Χ | (X응)<br>(X응)<br>(X응) | Χ | (X%)<br>(X%)<br>(X%) | X | (X%)<br>(X%)<br>(X%) | X | (X%)<br>(X%)<br>(X%) |
| | XXXXXXX | XXXX<br>XXXX<br>XXXX | Χ | (X%)<br>(X%)<br>(X%) | | (X%)<br>(X%)<br>(X%) | | (X%)<br>(X%)<br>(X%) | Χ | (X%)<br>(X%)<br>(X%) | X | (X%)<br>(X%)<br>(X%) | X | (X%)<br>(X%)<br>(X%) |

\_\_\_\_\_\_

 $\label{eq:product A = myblu^m closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 2.5 \%$ 

 $\label{eq:product B} \textit{Product B} = \textit{myblu}^{\text{TM}} \textit{ closed system with CF Cosmic Fog Tobacco Chill flavor, nicotine salt liquid 4.0\% } \\$ 

Product C = myblu™ closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 2.5 %

Product D =  $myblu^{mm}$  closed system with CF Cosmic Fog Honeymoon flavor, nicotine salt liquid 4.0%

Product E = Subject's usual brand combustible cigarette

Product F = JUUL® system with Virginia Tobacco Flavor JUUL pod, 5.0% nicotine

Program: /AAXXXXX/ECR/sas prg/stsas/tab programname.sas DDMMMYYYY HH:MM

#### Clinical Study Report No. CA22747

Table 14.3.1.1 Product Use-emergent Adverse Event Frequency by Study Product - Number of Subjects Reporting the Event
(% of Subjects Who Used Study Product) (Safety Population)

#### Product Trial# Adverse Event\* Number of Subjects Who Received Study Product XX(100%) Number of Subjects With Adverse Events X(X%) X(X%)Eve disorders $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ Vision blurred $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8) X(X_8)$ Gastrointestinal disorders $X(X_8)$ X(X%)X(X%)X( Dyspepsia X%) X ( X%) X ( X%) X ( X%) $X(X_8) X(X_8)$ Nausea $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8) X(X_8)$ Musculoskeletal and connective tissue $X(X\%) \times (X\%) \times (X\%) \times (X\%) \times (X\%) \times (X\%)$ $X(X_8)$ $X(X_8)$ disorders Back pain X(X%) $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ X%) $X(X_8)$ $X(X_8)$ X(X%)X( X%) X(X%) X(X%)X( $X(X_8)$ $X(X_8)$ Muscle cramps Musculoskeletal pain $X(X^{\circ})$ $X(X^{\circ})$ $X(X^{\circ})$ $X(X^{\circ})$ $X(X^{\circ})$ $X(X^{\circ})$ X(X) X(X) $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ Nervous system disorders $X(X_8)$ $X(X_8)$ Headache NOS $X(X_8)X(X_8)$ X%) X(X%) X(X%) X(X%) $X(X_8)$ $X(X_8)$ Χ( X%) Reproductive system and breast disorders X(X%) X(X%) X(X%) X(X%) X(X%) X(X%) $X(X_8)$ $X(X_8)$ Vaginal discharge $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8)$ $X(X_8) X(X_8)$

Note: \* Adverse events are classified according to MedDRA Version 21.0.

Product X: < >

Program: /CAXXXX/sas\_prg/stsas/tab cdash\_tblae1a\_auto.sas DDMMMYYYY HH:MM

<sup>#</sup> Only include the adverse events occurred during the product trial period.

<sup>^</sup> Adverse events occurred during the product trial period are excluded from Overall summary.

### Clinical Study Report No. CA22747


Table 14.3.1.2 Product Use-emergent Adverse Event Frequency by Study Product - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

| Adverse Event* | | Product<br>Trial# | | А | | В | | С | | D | E<br>XX (100%) | | F<br>XX(100%) | | Overall^<br><br>XX(100%) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of Adverse Events | XX (2 | L00%) | XX (100% | | XX(100%) | | XX(100%) | | XX (100%) | | | | | | | |
| Eye disorders | X ( | X%) | X ( | X%) | X ( | X%) | X ( | X%) | X ( | X%) | X ( | X%) | Х( | X%) | Х ( | <br>X%) |
| Vision blurred | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Gastrointestinal disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Dyspepsia | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Nausea | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Musculoskeletal and connective tissue | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| disorders | | | | | | | | | | | | | | | | |
| Back pain | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Muscle cramps | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Musculoskeletal pain | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Nervous system disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Headache NOS | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Reproductive system and breast disorders | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) |
| Vaginal discharge | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | Х ( | X%) | X ( | X%) | Х ( | X%) |

Note: \* Adverse events are classified according to MedDRA Version 21.0.

Product X: < >

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tblae2a\_auto.sas DDMMMYYYYY HH:MM

<sup>#</sup> Only include the adverse events occurred during the product trial period.

<sup>^</sup> Adverse events occurred during the product trial period are excluded from Overall summary.

#### Clinical Study Report No. CA22747


Table 14.3.1.3 Adverse Event Frequency by Study Product, Intensity, and Relationship to Study Product
- Number of Subjects Reporting Events (Safety Population)

| | 044 | Number of | | Intens | sity | Relationship to Study Product | | |
|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Study<br>Product<br> | Subjects with Adverse Events | Mild M | oderate | Severe | Unrelated | Possibly | Probably |
| Abdominal pain | X | X | X | X | X | X | X | X |
| Constipation | X | X | X | X | X | X | X | X |
| Dry throat | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X |
| Product Trial# | | X | X | X | X | X | X | X |
| Study Product A | | X | X | X | X | X | X | X |
| Study Product B | | X | X | X | X | X | X | X |
| Study Product C | | X | X | X | X | X | X | X |
| Study Product D | | X | X | X | X | X | X | X |
| Study Product E | | X | X | X | X | X | X | X |
| Study Product F | | X | X | X | X | X | X | X |
| Overall^ | | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.0.

When a subject experienced the same AE at more than one level of intensity during a product use period, only the most severe one was counted.

When a subject experienced the same AE at more than one level of product relationship during a product use period, only the one most closely related to study product was counted.

Product X: < >

Program: /CAXXXXX/sas prg/stsas/tab cdash tblae3a auto.sas DDMMMYYYY HH:MM

<sup>#</sup> Only include the adverse events occurred during the product trial period.

<sup>^</sup> Adverse events occurred during the product trial period are excluded from Overall summary.

Clinical Study Report No. CA22747

Table 14.3.2.1 Serious Adverse Events


There were no serious adverse events recorded during the study

Program: /CAXXXXX/sas\_prg/stsas/tab cdash\_tblae\_ser.sas DDMMMYYYY HH:MM

#### Clinical Study Report No. CA22747

#### Tables 14.3.4.1 to 14.3.4.3 will be in the following format:

Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry (Safety Population)

| Subject<br>Number | _ | Study<br>Period | Day | Hour | Date | Time | Parameter1<br><range><br/>(Unit)</range> | Parameter2<br><range><br/>(Unit)</range> | Parameter3<br><range><br/>(Unit)</range> | Parameter4<br><range><br/>(Unit)</range> | Parameter5<br><range><br/>(Unit)</range> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | XX/X | Screen<br>X | X | xx.xx | DDMMYYYY<br>DDMMYYYY | | | XX IN | | XX LYR+ | XX HN |

Note: # Age is calculated from the date of the first product use. F = Female, M = Male

H = Above normal range, L = Below normal range

Computer: N = Not clinically significant, Y = Clinically significant

PI Interpretation: - = Not clinically significant, R = Recheck requested, ^ = Will be retested later, + = Clinically significant

Programmer Notes: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Tables 14.3.4.2 and 14.3.4.3 will resemble 14.3.4.1.

Programmer Notes: Clinically significant lab values generally will be captured as AEs, some of which the PI may indicate in Appendix 16.2.8.1.5 lab comments (as per GPG.03.0028 sections 2.9 and 2.10). Derive an additional CS flag for PI flag (+) based on positive comments (i.e. CS/Clinically Significant). Present this derived 4<sup>th</sup> column in all tables, and list only subjects/tests which are PI-determined clinically significant lab values in Table 14.3.4.4.

Program: /CAXXXX/sas prg/stsas/tab PROGRAMNAME.sas DDMMYYYY HH:MM

#### Clinical Study Report No. CA22747

#### Table 14.3.4.4 will be in the following format:

Table 14.3.4.4 Clinically Significant Values and Recheck Results (Safety Population)

| Subject Age#/<br>Number Sex | Study<br>Period | Day Hour | Date | Time | Department | Test | Res | ult | Normal Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|
| X XX/X | Х | | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX | XXX | HYR+ | X - X | mg/dL |

< All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table. >

Note: # Age is calculated from the date of the first product use. F = Female, M = Male H = Above normal range

Computer: Y = Clinically significant

PI Interpretation: R = Recheck requested, + = Clinically significant

Program: /CAXXXXX/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: If no event meet this criteria then include a statement as follows: "There were no clinical laboratory results documented as clinically significant by the PI."

#### Tables 14.3.5.2 and 14.3.5.3 will resemble Table 14.3.5.1

Table 14.3.5.1 Clinical Laboratory Summary - Serum Chemistry (Safety Population)

| | | m : | | Product | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (units) | Normal<br>Range | Time<br>Point | Statistic | A | В | C | D | E | F |
| Testname (unit) | < - ># | Screen | n | X | X | Х | Х | Х | Х |
| | | | Mean | X.X* | X.X | X.X* | X.X | X.X* | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | | Check-in | n | X | X | X | X | Х | X |
| | | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |

Note: # = Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

<sup>\*</sup> Above Normal Range, ^ Below Normal Range Product X: <>

<sup>&</sup>lt; Similar for remaining laboratory tests. >

### Clinical Study Report No. CA22747

Page 1 of X Table 14.3.5.4 Vital Sign Summary Vital Sign Summary at Screening, Check-in, and Prior to Discharge (Safety Population)

| | | | Product | | | | | |
|---|---|---|---|---|---|---|---|---|
| Vital Sign (units) | Time<br>Point | Statistic | А | В | С | D | E | F |
| Testname (unit) | Screen | n | X | Х | Х | Х | Х | Х |
| | | Mean | X.X* | X.X | X.X* | X.X | X.X* | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX |
| | Check-in | n | Х | Х | Х | Х | X | Х |
| | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX | XX | XX | XX |
| | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX | XX | XX | XX |

< Similar for remaining vital signs and time points. >

Note: Product X : < >

Program: /CAXXXXX/ECR/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

Clinical Study Report No. CA22747

#### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final report. These listings will be generated off of the SDTM Version 1.4. All listings will be presented in Courier New size font 9.

### Clinical Study Report No. CA22747


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Gender | Age Category | Normal Range | Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name | | | XX - XX | units |
| 1 | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| Hematology | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| 31 | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Leftrightarrow$ | $\Diamond$ | XX - XX | units |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Similar for remaining Laboratory Groups and Test Names.

### Clinical Study Report No. CA22747


Appendix 16.2.1 Subject Discontinuation

| Subject<br>Number | Date | Product | Completed<br>Study? | Reason for Discontinuation Specify |
|---|---|---|---|---|
| X | DDMMYYYY | X | Yes | |
| X | DDMMYYYYY | X | Yes | |
| X | DDMMYYYYY | X | Yes | |
| X | DDMMYYYYY | X | Yes | |
| X | DDMMYYYYY | X | No | Personal Reason |
| X | DDMMYYYYY | X | Yes | |
| X | DDMMYYYYY | X | Yes | |
| X | DDMMYYYY | X | Yes | |

Note: Product X: < >

### Clinical Study Report No. CA22747


Appendix 16.2.4.1.1 Subject Information (Safety Population)

| Subje | Informed<br>ect Consent | Protocol | Pandomization | Randomization | Study | Subject<br>Previously | Previous<br>Subject | Re-coi | nsent |
|---|---|---|---|---|---|---|---|---|---|
| Numbe | | Version | Number | Date | Product | Screened? | Number | Version | Date |
| | X DDMMYYYY | X | XX | DDMMYYYY | X | XX | | | |
| | X DDMMYYYYY | X | XX | DDMMYYYYY | X | XX | | | |

\_ \_ \_

Note: Product X: < >

### Clinical Study Report No. CA22747


Appendix 16.2.4.1.2 Demographics (Safety Population)

| Subject<br>Number | Age<br>(yrs) | Sex | Race | Reproductive<br>Status | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) |
|---|---|---|---|---|---|---|---|---|
| X | XX | XXXX | XXXXXXXXX | XXXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX |
| X | XX | XXXX | XXXXXXXX | XXXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX |

### Clinical Study Report No. CA22747


Appendix 16.2.4.1.3 Additional Demographics Questionnaire (Safety Population)

| Subject<br>Number | Income* | Grade* | Marital Status | Identity* |
|-------------------|-----------|-------------|----------------|-------------|
| X | XXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXX |
| X | XXXXXXXX | XXXXXXXXXX | XXXXXXXXXX | XXXXXXXXXX |
| X | XXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXX | XXXXXXXXXXX |

Note: \* Income = What was your annual household income from all sources over the past year? Grade = What was the highest grade or year of school you completed? Identity = Which of the following options do you identify with?

## Clinical Study Report No. CA22747

Appendix 16.2.4.2.1 Physical Examination - Full (Safety Population)


| Subject<br>Number | Study<br>Visit | Date | Was PE<br>Performed? | Reason for<br>Not Done | Body System | If Other,<br>Specify | Result | Specify if Abnormal or Not Done |
|---|---|---|---|---|---|---|---|---|
| Х | Screening | DDMMYYYY | XXX | | XXXXXXXX | | XXXX | |

### Clinical Study Report No. CA22747

Appendix 16.2.4.2.2 Physical Examination - Symptom-driven (Safety Population)

| Page 1 | of | Σ |
|--------|----|---|
|--------|----|---|

| Subject<br>Number | Study<br>Visit | Date | Report<br>Symptom? | Was PE<br>Performed? | Reason for<br>Not Done | Abnormal Findings? | Body System | If Other,<br>Specify | Result | Specify if Abnormal |
|---|---|---|---|---|---|---|---|---|---|---|
| | VVV | | | YYY | | | | | | |

### Clinical Study Report No. CA22747

Appendix 16.2.4.3 Medical and Surgical History (Safety Population)

| Subject<br>Number | | Study<br>Visit | MH<br>Number | Category | Body Sy | rstem | Report term | Onset<br>Date | Ongoing | End<br>Date |
|---|---|---|---|---|---|---|---|---|---|---|
| X | XXX | Screening | X | XXXXXXX | XXXXXXX | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | Yes | |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747


Appendix 16.2.4.4.1 Tobacco/Nicotine Product Use History Questionnaire (Safety Population)

| Subject | Study | Questionnaire | |
|--------------|-----------|---------------|-----------|
| Number Visit | | Completed? | Date |
| X | Screening | XXX | DDMMYYYYY |

## Clinical Study Report No. CA22747


Appendix 16.2.4.4.2 Smoking History (Safety Population)

| Subject | Study | Number of Years | Average Number of Cigarettes |
|---------|-----------|--------------------|------------------------------|
| Number | Visit | Smoked Cigarettes? | Smoked During the Past Year |
| Х | Screening | XXX | XX |

### Clinical Study Report No. CA22747

Appendix 16.2.4.4.3 Usual Brand Documentation (Safety Population)

| Subject<br>Number | Study<br>Visit | Usual Brand<br>Changed?* | Color<br>Photocopy?* | Brand | If Other, Specify | Brand Style | Flavor | Length |
|---|---|---|---|---|---|---|---|---|
| X | XXXXX | XXXXXX | XXX | XXXXXX | | XXXXXXXX | XXX | XXXXX |

Note: \* Usual Brand Changed? = Has subject's usual brand changed since last reported?

\* Color Photocopy? = Was a color photocopy of subject's usual brand cigarette package obtained?

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

## Clinical Study Report No. CA22747

Appendix 16.2.5.1 Inclusion / Exclusion Criteria Not Met (Safety Population)

| Subject<br>Number | Study<br>Visit | Did subject meet all eligibility criteria? | Criterion<br>Identifier | Inclusion/Exclusion<br>Category | Did the Subject<br>Enroll? |
|---|---|---|---|---|---|
| X | Screening | No | EXCLUSION X | XXXXXXXXXXXXXXX XXXX | XXX |
| X | Screening | Yes | | | |
| X | Screening | Yes | | | |

Program: /CAXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMYYYYY HH:MM

### Clinical Study Report No. CA22747


Appendix 16.2.5.2.1 myblu™ Product Preference Questionnaire (Safety Population)

| Subject<br>Number | | Product | Rank |
|-------------------|-----|-------------------------------|------|
| X | XXX | Tobacco Chill - low nicotine | X |
| | | Tobacco Chill - high nicotine | X |
| | | Honeymoon - low nicotine | X |
| | | Honeymoon - high nicotine | X |

## Clinical Study Report No. CA22747


Appendix 16.2.5.2.2 Product Selection (Safety Population)

| Subject<br>Number | _ | Initial Product<br>Selected | Switch?* | Product Selected<br>To Continue |
|---|---|---|---|---|
| X | XXX | X | XXX | × |

Note: Product X: < >

\* = Indicate how subject would like to continue

### Clinical Study Report No. CA22747


Appendix 16.2.5.2.3 Staff-Recorded In-Clinic Product Use (Safety Population)

| Subject<br>Number | Study<br>Day | Product | Date | Number of<br>Cigarettes<br>Smoked | Number of New<br>New Pods<br>Started | FAS<br>Flag | PP28/29<br>Flag | PP56/57<br>Flag | |
|---|---|---|---|---|---|---|---|---|---|
| X | X | X | DDMMYYYY | X | X | X | X | X | _ |

Note: . = Missing or not reportable, NA = Not applicable, Y = Included, N = Excluded Product X = <  $\,>\,$ 

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: Puff and cartridge categories apply only to subjects using myblu™ products

### Clinical Study Report No. CA22747


#### Appendix 16.2.5.2.4 Self-Reported Product Use (Safety Population)

| Subject<br>Number | Study<br>Day | Product | Date | Number of<br>Cigarettes<br>Smoked | Number of New<br>New Pods<br>Started | Take More Than<br>50 Puffs From<br>myblu™ Today? | FAS PP28/29<br>Flag Flag | , - | |
|---|---|---|---|---|---|---|---|---|---|
| Х | X | Х | DDMMYYYY | X | X | X | X | X X | ζ |

Note: . = Missing or not reportable, NA = Not applicable, Y = Included, N = Excluded Product X = < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: Puff and cartridge categories apply only to subjects using myblu™ products
### Clinical Study Report No. CA22747

Page 1 of X Appendix 16.2.5.2.5 Product Use - Nicotine PK Assessment (Safety Population)

| | | | Is Session Data<br>Available? | | | | | | | | Number of<br>Puffs Taken |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Х | -<br>XXX | Х | XXXX | DDMMYYYY | HH:MM | X<br>X<br>X | X.XXXX<br>X.XXXX<br>X.XXXX | HH:MM | X.XXXX<br>X.XXXX<br>X.XXXX | HH:MM<br>HH:MM | XX<br>XX<br>XX |

Note: Product X: < >

### Clinical Study Report No. CA22747


Appendix 16.2.5.3.1 Pharmacokinetics Blood Sampling (Safety Population)

| Subject<br>Number | | Study<br>Product | Was Blood Sample<br>Collected? | Bioassay | Scheduled Timepoint | Date | Actual<br>Time | Comments |
|---|---|---|---|---|---|---|---|---|
| X | X | X | XXX | XXXXX | XXXXXXXXXXXXXXXXXX | DDMMYYYY | HH:MM | |
| | | | | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYYY | HH:MM | |
| | | | | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYYY | HH:MM | |
| | | | | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | HH:MM | |

Note: Product X: < >

### Clinical Study Report No. CA22747


Appendix 16.2.5.3.2 24-Hour Urine Collection (Safety Population)

| | | Study<br>Product | Was Urine Sample<br>Collected? | Reason for<br>Not Done | | Start<br>Time | End<br>Date | | Total Urine<br>Weight (g) | 2 | Reason for<br>Missing Void |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | X | X | XXX | | DDMMMYYYY | HH:MM | DDMMYYYY | HH:MM | XXXX | XX | |

Note: Product X: < >

### Clinical Study Report No. CA22747

Page 1 of X Appendix 16.2.5.3.3 24-Hour Urine Collection - Pod Weight Documentation (Safety Population) (Safety Population)

| | | | Number of Pods Used During<br>24-hour Urine Collection | Pod<br>Number | Pod Starting<br>Weight (g) | Pod End<br>Weight (g) |
|---|---|---|---|---|---|---|
| X | Х | X | XXX | X | X.XXXX | X.XXXX |
| | | | | X | X.XXXX | X.XXXX |
| | | | | X | X.XXXX | X.XXXX |

Note: Product X: < >

### Clinical Study Report No. CA22747

Page 1 of X Appendix 16.2.5.3.4 Carboxyhemoglobin Blood Collection (Safety Population)

| _ | | Study<br>Product | Were Blood Sample for COHb Collected? | Reason for<br>Not Done | Collection<br>Date | Collection<br>Time | |
|---|---|---|---|---|---|---|---|
| X | X | Х | XXX | | DDMMYYYY | HH:MM | _ |

### Clinical Study Report No. CA22747


Appendix 16.2.5.3.5 Biomarkers and Bio-Banking Blood Collection (Safety Population)

| _ | | Study<br>Product | Were Blood Sample for Biomarkers and Biobanking Collected? | Reason for<br>Not Done | Collection<br>Date | Collection<br>Time |
|---|---|---|---|---|---|---|
| X | X | X | XXX | | DDMMYYYY | HH:MM |

### Clinical Study Report No. CA22747

Appendix 16.2.5.4 Prior and Concomitant Medications (Safety Population)

| Subject<br>Number | | Study Any<br>Product Med? | | Dosage | Route | Start<br>Date | Stop<br>Date | Frequency | MH<br>/ Indication Term | AE<br>n Term | Ongoing? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| X | XXXX | X XXX | XXXXXXXXXXX<br>(XXXXXXXXXXXX) | 620 mg O | RAL | DDMMYYYY | DDMMYYYY | Once | Toothache | | No |

Note: \* Concomitant medications are coded with WHO Dictionary Version DDMMMYYYY. Product X: < >

Program: /CAXXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMYYYYY HH:MM

### Clinical Study Report No. CA22747

#### Appendices for blood biomarkers will have the following format:

Appendix 16.2.6.2.1 Whole Blood COHb (Outcomes Population)


| Subject<br>Number | Product | Planned Visit | Study<br>Day | COHb<br>(% Saturation) | Change From Baseline (% Saturation) | % Change From<br>Baseline | FAS<br>Flag | PPS<br>5/6<br>Flag | PPS<br>29/30<br>Flag | PPS<br>59/60<br>Flag |
|---|---|---|---|---|---|---|---|---|---|---|
| X | X | Day -1 | -X | X.X | NA | NA | Y | X | X | Х |
| | | Day 5 | X | X.X | X.X | XX.XX | Y | X | X | X |
| | | Day 29 | XX | X.X | X.X | XX.XX | Y | NA | X | X |
| | | Day 59 | XX | X.X | X.X | XX.XX | Y | NA | NA | X |

Note: Product X: < >

### Clinical Study Report No. CA22747

#### Appendices for urine biomarkers will have the following format:

Appendix 16.2.6.2.2 Urine NNAL (Outcomes Population)


| Subject | Droduct | | Creatinine | NNAL | | (ng/g | Cr) | Weight | Excreted | | eted | | PPS<br>5/6 | PPS<br>29/30 | PPS<br>59/60 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Product | Day | (mg/L)<br> | (pg/mL) | (ng/g Cr) | | % Change | (g)<br> | (ng/24hrs)<br> | | % Change<br> | riag | riag | Flag<br> | Flag |
| 03-0010 | X | <b>-</b> X | XXX | XXX | XXX | NA | NA | XXXX | XXXX | NA | NA | Y | Y | Y | Y |
| | | X | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XXX | XXX | Y | Y | Y | Y |
| | | XX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XXX | XXX | Y | N | Y | Y |
| | | XX | XXX | XXX | XXX | XXX | XXX | XXXX | XXXX | XXX | XXX | Y | N | N | Y |

Note: Product X: < >

#### Clinical Study Report No. CA22747


Appendix 16.2.6.3.1 PSCDI, PSECDI Questionnaire (ITT Population)

- 1. How many cigarettes [times] per day do you usually smoke [use your electronic cigarette]? ([assume that one "time" consists of around 15 puffs or lasts around 10 minutes]) (Scoring: 0-4 times/day = 0, 5-9 = 1, 10-14 = 2, 15-19 = 3, 20-29 = 4, 30+ = 5)
- 2. On days that you can smoke [use your electronic cigarette] freely, how soon after you wake up do you smoke your first cigarette of the day [first use your electronic cigarette]? (Scoring: 0-5 mins = 5, 6-15 = 4, 16-30 = 3, 31-60 = 2, 61-120 = 1, 121+ = 0)
- 3. Do you sometimes awaken at night to have a cigarette [use your electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 4. If yes, how many nights per week do you typically awaken to smoke [use your electronic cigarette]? (Scoring: 0-1 nights = 0, 2-3 nights = 1, 4+ nights = 2)
- 5. Do you smoke [use an electronic cigarette] now because it is really hard to quit? (Scoring: Yes = 1, No = 0)
- 6. Do you ever have strong cravings to smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 7. Over the past week, how strong have the urges to smoke [use an electronic cigarette] been? (Scoring: None/Slight = 0, Moderate/Strong= 1, Very Strong/Extremely Strong = 2)
- 8. Is it hard to keep from smoking [using an electronic cigarette] in places where you are not supposed to? (Scoring: Yes = 1, No = 0)

When you haven't used tobacco [an electronic cigarette] for a while or when you tried to stop smoking [using]...

- 9. Did you feel more irritable because you couldn't smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 10. Did you feel nervous, restless, or anxious because you couldn't smoke [use an electronic cigarette]? (Scoring: Yes = 1, No = 0)
- 11. Total scoring: 0 3 = not dependent, 4 8 = low dependence, 9 12 = medium dependence, 13+ = high dependence.

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### Nerudia Ltd.

#### *my*blu E-cigarettes

### Clinical Study Report No. CA22747

Appendix 16.2.6.3.2 PSCDI, PSECDI Questionnaire Responses (ITT Population)

| Subject | | Time | | | | | | | Questi | on | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Product | Point | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | Total Score |
| XXXXXX | X | XXXX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |

Note: Product X: < >

Refer to Appendix 16.2.6.3.1 for the description of questions.

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747


Appendix 16.2.6.4.1 Cough Questionnaire (ITT Population)

- 1. Did you have a cough during the last 5 days?
- 2. How would you rate the intensity of your cough during the last 5 days?
- 3. How often did you cough up phlegm during the last 5 days?
- 4. How often did your cough disturb your sleep during the last 5 days?
- 5. How often did you have coughing bouts during the day, during the last 5 days?

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

### Nerudia Ltd.

### *my*blu E-cigarettes

### Clinical Study Report No. CA22747

Appendix 16.2.6.4.2 Cough Questionnaire Responses (ITT Population)


| Subject<br>Number | Product | Time<br>Point | 1 | 2 | Question<br>3 | 4 | 5 |
|---|---|---|---|---|---|---|---|
| XXXXXX | X | XXXX | XXXXXXXXX | XXXXXXXXX | XXXXXXXXXXXX | x xxxxxxxxx | XXXXXXXXXXX |

Note: Product X: < >

Refer to Appendix 16.2.6.4.1 for the description of questions.

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747


Appendix 16.2.6.5.1 MTWS-R Questionnaire (ITT Population)

Please rate yourself for the period of the last 24 hours.

- 1. Angry, irritable, frustrated
- 2. Anxious, nervous
- 3. Depressed mood, sad
- 4. Difficulty concentrating
- 5. Increased appetite, hungry, weight gain
- 6. Insomnia, sleep problems, awakening at night
- 7. Restless
- 8. Desire or craving to smoke

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Nerudia Ltd.

#### myblu E-cigarettes

#### Clinical Study Report No. CA22747

Appendix 16.2.6.5.2 MTES-R Questionnaire Responses (ITT Population)

 Subject
 Time
 Question

 Number
 Product
 Point
 1
 2
 3
 4
 5
 6
 7
 8
 Total Score

 XXXXXX
 X
 XXXXXX
 X

Note: Product X: < >

Scale: 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Refer to Appendix 16.2.6.5.1 for the description of questions.

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

### Clinical Study Report No. CA22747

Appendix 16.2.6.6.1 QSU-brief Questionnaire (ITT Population)


1. <> 2. <>

3. < >

4. < > 5. <>

6. < >

7. <>

8. < >

9. <>

10. <>

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

### Nerudia Ltd.

#### myblu E-cigarettes

#### Clinical Study Report No. CA22747

Appendix 16.2.6.5.2 MTES-R Questionnaire Responses (ITT Population)

Note: Product X: < >

Scale: 1 = Strongly disagree, 7 = Strongly agree

Factor 1 (anticipation of pleasure from smoking): average of items 1, 3, 6, 7, and 10.

Factor 2 (relief of nicotine withdrawal): average of items 2, 4, 5, 8, and 9.

Refer to Appendix 16.2.6.6.1 for the description of questions.

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### Clinical Study Report No. CA22747


Appendix 16.2.6.7.1 PES Questionnaire (ITT Population)

- 1. Was it satisfying?
- 2. Did it taste good?
- 3. Did you enjoy the sensations in your mouth?
- 4. Did it calm you down?
- 5. Did it make you feel more awake?
- 6. Did it make you feel less irritable?
- 7. Did it help you concentrate?
- 8. Did it reduce your hunger for food?
- 9. Did it make you dizzy?
- 10. Did it make you nauseous?
- 11. Did it immediately relieve your craving for a cigarette?
- 12. Did you enjoy it?
- 13. Did it relieve withdrawal symptoms?
- 14. Did it relieve the urge to smoke?
- 15. Was it enough nicotine?
- 16. Was it too much nicotine?
- 17. Was it easy to use?
- 18. Were there bothersome side effects?
- 19. Were you comfortable using the product in public?
- 20. Did you still have a craving for a cigarette after using the product?
- 21. Are you concerned that you would become dependent on this product?

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Nerudia Ltd.

#### *my*blu E-cigarettes

#### Clinical Study Report No. CA22747

Appendix 16.2.6.7.2 PES Questionnaire Responses (ITT Population)

Subject Time ----- Ouestion -----Number Product Point Χ XXXXXX XXXX

Note: Product X: < >

Scale: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely Refer to Appendix 16.2.6.7.1 for the description of questions.

Program: /CAXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### Clinical Study Report No. CA22747

Appendix 16.2.6.7.3 PES Questionnaire Subscales (ITT Population)

| Subject | | Time | | Questio | n | |
|---|---|---|---|---|---|---|
| Number | Product | Point | Satisfaction | Psychological Reward | Aversion | Relief |
| | v | VVVV | | v | Y | |

Note: Product X: < >

"Satisfaction" (items 1, 2, 3, and 12);
"Psychological Reward" (items 4 through 8);
"Aversion" (items 9, 10, 16, and 18);
"Relief" (items 11, 13, 14, 15, and reversed for item 20)

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

### Clinical Study Report No. CA22747

Appendix 16.2.6.8 Product Liking Questionnaire Responses (ITT Population)


| Subject<br>Number | Product | Time<br>Point | Question | VAS Score |
|-------------------|---------|---------------|----------|-----------|
| XXXXXX | X | XXXX | | XX |

Note: Product X: < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747

Appendix 16.2.6.9 Future Intent to Use Questionnaire Responses (ITT Population)

Subject Time Number Product Point Question VAS Score XXXXXX XXXX XX XX XXXX XX XX

Note: Product X: < >

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYY HH:MM

### Clinical Study Report No. CA22747

Page 1 of X Appendix 16.2.6.10 Product and Health Effect Perceptions Questionnaire Responses (ITT Population)

| Subject<br>Number | Product | Time<br>Point | Question | VAS Score |
|---|---|---|---|---|
| XXXXXX | Χ | XXXX | | XX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX |
| | | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX |

Note: Product X: < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

#### Clinical Study Report No. CA22747


Appendix X Urge to Smoke Assessments (PK Population)

| Subject<br>Number | Product | Time<br>Point | Question | VAS Score |
|---|---|---|---|---|
| XXXXXX | X | XXXX<br>XXXX | How strong is your urge to smoke right now? How strong is your urge to smoke right now? | XX<br>XX |

Note: Product X: < >

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programmer Note: This listing also can be presented as horizontal format. It will only be presented for the sub-study.

#### Clinical Study Report No. CA22747


#### Appendix 16.2.7.1.1 Adverse Events (I of II) (Safety Population)

| | | | | | | Onset | | Resolved | | Duration |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Study | | | | | | | | |
| Number | Visit | Product | UE?^ | Adverse Event* | Preferred Term | Date | Time | Date | Time | (DD:HH:MM) |
| 1 | X | X | Yes | XXXXXXXXXXXX | XXXXXXXXXX XXXXXXX | DDMMYYYYY | X:XX | DDMMYYYYY | X:XX | XX:XX:XX |

Note: & = Abbreviation for study product use-emergent (UE),

\* = Adverse events are classified according to the MedDRA Version XX.X.

Product X: < >

### Clinical Study Report No. CA22747


Appendix 16.2.7.1.2 Adverse Events (II of II) (Safety Population)

| | | | | Onset | | | | | | Relation-<br>ship to | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | | Study<br>Product | Adverse<br>Event | Date | Time | Freq | Severity | Ser* | Outcome | Study<br>Product | Action |
| 1 | XXX | X | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYYY | X:XX | Inter | . Mild | XXX | Resolved | XXXXXXXX | None |

Note: Ser\* represents Serious event.

Freq represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Product X: < >

### Clinical Study Report No. CA22747


#### Appendix 16.2.7.2 Adverse Event Preferred Term Classification (Safety Population)

| | | | | | | Unset | |
|---|---|---|---|---|---|---|---|
| Subject | Study | Study | Adverse | | | | |
| Number | Visit | Product | Event | Preferred Term | Body System | Date | Time |
| 1 | X | X | XXXXXXX XXXXX XXXX XXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY | X:XX |

Note: \* = Adverse events are classified according to the MedDRA Version XX.X. Product X: < >

Clinical Study Report No. CA22747

#### Appendices 16.2.8.1.2 to 16.2.8.1.3 will have the following format.


Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Subject<br>Number | Age/<br>Sex | Study<br>Visit Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) | Parameter6<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|
| X | XX | Screening DDMMMYYYY XXXXXX DDMMMYYYY | | XX<br>XX | XX<br>XX | XX<br>XX | XX HN<br>XX HN | XX<br>XX |

Note: H = Above Reference Range, L = Below Reference Range PI flag: CS = Clinically significant, NCS = not clinically significant

 $\label{program: program: pro$ 

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study.

### Clinical Study Report No. CA22747


Appendix 16.2.8.1.4 Serology (Safety Population)

| Subject<br>Number | | Was the Sample<br>Collected? | Reason for Not Done | Date of Collection |
|---|---|---|---|---|
| X | Screening | XXX | | DD <b>MM</b> YYYY |

### Clinical Study Report No. CA22747

Appendix 16.2.8.1.5 Urine Drug Screen (Safety Population)


| | ct Study<br>r Visit | Was the Urine Sample<br>Collected? | Reason for<br>Not Done | Date of<br>Collection | Test Name | Result |
|---|---|---|---|---|---|---|
| X | Screening | XXX | | DDMMYYYY | XXXXXXX | XXXXXX |
| | | | | | XXXXXXX | XXXXXX |

### Clinical Study Report No. CA22747

Appendix 16.2.8.1.6 Alcohol Breath Test (Safety Population)


| _ | t Study<br>Visit | Was the Alcohol Breath<br>Test Performed? | Reason for<br>Not Done | Date of Test | Result |
|---|---|---|---|---|---|
| X | Screening | XXX | | DDMMYYYY | XXXXXX |

### Clinical Study Report No. CA22747

Appendix 16.2.8.1.7 Urine Cotinine Screen (Safety Population)

Subject Study Was the Urine Cotinine Reason for Date of
Number Visit Sample Collected? Not Done Collection Result

X Screening XXX DDMMYYYY XXXXXX

Program: /CAXXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747

Appendix 16.2.8.1.8 Pregnancy Test (Safety Population)


| _ | ct Study<br>Visit | Was the Pregnancy<br>Test Done? | Reason for<br>Not Done | Date of<br>Collection | Time | Category | Result |
|---|---|---|---|---|---|---|---|
| X | Screening | XXX | | DDMMYYYY<br>DDMMYYYYY | HH:MM | XXXXXX | XXXXXX |

### Clinical Study Report No. CA22747


Appendix 16.2.8.1.9 Serum FSH (Safety Population)

| Subject | 4 | Was the Sample | Reason for | Date of | Was Post-menopausal |
|---|---|---|---|---|---|
| Number | | Collected? | Not Done | Collection | Status Confirmed? |
| X | Screening | XXX | | DDMMMYYYY | XXX |

### Clinical Study Report No. CA22747


Appendix 16.2.8.2 Vital Signs (Safety Population)

| | | | | | | Blood Pressure (mmHg) | | Respir | - Temper- | - |
|---|---|---|---|---|---|---|---|---|---|---|
| Subjec | t Study | Was VS | Reason for | | | | Pulse | ation | ature | Weight |
| Number | Visit | Product Measured? | Not Done | Date | Time | Systolic/Diastolic | (bpm) | (rpm) | (℃) | (kg) |
| X | Screening | XXX | | DDMMYYYY | X:XX | XXX/ XX | XX | XX | XX.X | XXX.X |
| | X | X XXX | | DDMMMYYYY | XX:XX | XXX/ XX | XX | XX | XX.X | |

Note: Product X: < >

### Clinical Study Report No. CA22747

Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Page | 1 | of | Χ |
|------|---|----|---|
|------|---|----|---|

| | | | | | | | Heart | | | If Abnormal | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject St | - | ECG | Reason for | | | | Rate | PR | QRS | QΤ | QTcB* | | |
| Number Vi | sit | Done? | Not Done | Date | Time | Result | (bpm) | (msec) | (msec) | (msec) | (msec) | Specify | Action Taken |
| Y Scr | eenina | XXX | | | v•xx•xx | Normal | | XXX X | XX X | XXX X | XXX X | | |

Note: QTCB\* = QTc corrected using Bazett's correction.

### Clinical Study Report No. CA22747

Appendix 16.2.8.4 Carbon Monoxide Breath Test (Safety Population)

Subject Study Were Exhaled CO Reason for Number Visit Levels Measured Not Done Date Time Result (ppm)

X Screening XXX DDMMYYYY HH:MM XXX

Program: /CAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

### Clinical Study Report No. CA22747


Appendix 16.2.8.5 FeNO Measurement (Safety Population)

| Subjec<br>Number | t Study<br>Visit | Were FeNO Measurements Collected? | Reason for<br>Not Done | Date | Time | FeNO (ppb) | Comment |
|---|---|---|---|---|---|---|---|
| X | Screening | XXX | | DDMMYYYYY | HH:MM | XXX | |

### Clinical Study Report No. CA22747

Appendix 16.2.8.6 Spirometry (Safety Population)


| | | | | | | | FVC | | FEV1 | | FVC:FEV1 Ratio | | FEF 25-75% | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | t Study<br>Visit | Event* | Test<br>Done? | Reason for<br>Not Done? | Date | Time | M# (L) | P# (%) | M# (L) | P# (%) | <br>M# | P# | M# | P# |
| X | Screening | | XXX | | DDMMYYYY<br>DDMMYYYYY | | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Alb<br>Post | XXX | | DDMMYYYY | HH:MM<br>HH:MM | XX | XX | XX | XX | XX | XX | XX | XX |

Note: \* pre = pre-bronchodilator, Alb = Albuterol administration, post = post-bronchodilator # M = Measured, P = Predicted